CLINICAL TRIAL: NCT05289037
Title: Phase 2 Clinical Trial to Optimize Immune Coverage of SARS-CoV-2 Existing and Emerging Variants
Brief Title: COVID-19 Variant Immunologic Landscape Trial (COVAIL Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0004; 5UM1AI148684-03 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-03-21 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2022-10-03

CONDITIONS: COVID-19
Keywords: Adaptive; COVAIL; Covid-19; Multivalent; Omicron; SARS-CoV-2; Vaccine; Variants
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (17):
- Arm 01 (Experimental): mRNA-1273 administered through 0.2 mg/ml intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273; Other: Sodium Chloride, 0.9%
- Arm 02 (Experimental): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273.351; Biological: mRNA-1273.529; Other: Sodium Chloride, 0.9%
- Arm 03 (Experimental): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273.351; Biological: mRNA-1273.529; Other: Sodium Chloride, 0.9%
- Arm 04 (Experimental): 0.2 mg/ml of mRNA-1273.617.2 and 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273.529; Biological: mRNA-1273.617.2; Other: Sodium Chloride, 0.9%
- Arm 05 (Experimental): 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273.529; Other: Sodium Chloride, 0.9%
- Arm 06 (Experimental): 0.2 mg/ml of mRNA-1273.529 and mRNA-1273 0.2 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.529; Other: Sodium Chloride, 0.9%
- Arm 07 (Experimental): 500 mcg/mL of BNT162b2 (Wildtype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2
- Arm 08 (Experimental): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2 (B.1.1.529); Biological: BNT162b2 (B.1.351)
- Arm 09 (Experimental): 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2 (B.1.1.529)
- Arm 10 (Experimental): 500 mcg/mL of BNT162b2 (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2 (B.1.351)
- Arm 11 (Experimental): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Wildtype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2; Biological: BNT162b2 (B.1.351)
- Arm 12 (Experimental): 500 mcg/mL of BNT162b2 (Omicron) and 500 mcg/mL of BNT162b2 (Wildtype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Biological: BNT162b2; Biological: BNT162b2 (B.1.1.529)
- Arm 13 (Experimental): 500 mcg/mL CoV2 preS dTM-AS03 [D614] (prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Drug: AS03; Biological: CoV2 preS dTM/D614
- Arm 14 (Experimental): 500 mcg/mL CoV2 preS dTM-AS03 [B.1.351] (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Drug: AS03; Biological: CoV2 preS dTM [B.1.351]
- Arm 15 (Experimental): 500 mcg/mL CoV2 preS dTM-AS03 [D614 + B.1.351] (prototype + Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  Interventions: Drug: AS03; Biological: CoV2 preS dTM/D614+B.1.351
- Arm 16 (Experimental): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.1) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years; ( 45% in > / = 49 years) N=100
  Interventions: Biological: BNT162b2 bivalent (wildtype and Omicron BA.1)
- Arm 17 (Experimental): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years; ( 45% in > / = 49 years) N=100
  Interventions: Biological: BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5)

INTERVENTIONS:
Drug: AS03 — AS03 oil-in-water emulsion adjuvant.
  Arms: Arm 13; Arm 14; Arm 15
Biological: BNT162b2 — A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2.
  Arms: Arm 07; Arm 11; Arm 12
Biological: BNT162b2 (B.1.1.529) — A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Arms: Arm 08; Arm 09; Arm 12
Biological: BNT162b2 (B.1.351) — A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.
  Arms: Arm 08; Arm 10; Arm 11
Biological: BNT162b2 bivalent (wildtype and Omicron BA.1) — A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer. Contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.1 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2.
  Arms: Arm 16
Biological: BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5) — A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer. Contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2.
  Arms: Arm 17
Biological: CoV2 preS dTM [B.1.351] — Is a liquid formulation made of recombinant protein placed in a formulation buffer that contains the spike protein sequence of the B.1.351 (Beta) variant SARS-CoV-2 strain.
  Arms: Arm 14
Biological: CoV2 preS dTM/D614 — Is a liquid formulation made of recombinant protein placed in a formulation buffer. The antigen solution contains the spike protein sequence of the ancestral strain of SARS-CoV-2.
  Arms: Arm 13
Biological: CoV2 preS dTM/D614+B.1.351 — Is a liquid formulation made of recombinant protein placed in a formulation buffer contains the spike protein sequences of the ancestral and B.1.351 (Beta) variant SARS-CoV-2 strains
  Arms: Arm 15
Biological: mRNA-1273 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
  Arms: Arm 01; Arm 06
Biological: mRNA-1273.351 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike (S) protein of the B.1.351 variant SARS-CoV-2 strain.
  Arms: Arm 02; Arm 03
Biological: mRNA-1273.529 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Arms: Arm 02; Arm 03; Arm 04; Arm 05; Arm 06
Biological: mRNA-1273.617.2 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.617.2 (Delta) variant SARS-CoV-2 strain.
  Arms: Arm 04
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection
  Arms: Arm 01; Arm 02; Arm 03; Arm 04; Arm 05; Arm 06

SUMMARY:
This phase 2 clinical trial will evaluate the safety and immunogenicity of additional doses of prototype and variant (alone or in combination) vaccine candidates in previously vaccinated participants with or without prior severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and will evaluate innate, cellular, and humoral immune responses to inform on how to shift the immune response to cover new variants as they emerge. A randomized open-label, non-placebo controlled, multi-site, multi-stage clinical trial in individuals, 18 years of age and older, who are in a stable state of health, has received a complete authorized/approved vaccine series (primary series + booster either with homologous or heterologous vaccine products) >/ = 16 weeks prior to enrollment. Subjects will be stratified by i) age (18-64 years and = 65 years of age) (however arms 16 and 17 or stage 4 will only enroll participants between the ages of 18-49 years) and ii) history of confirmed prior SARS-CoV-2 infection, and randomly assigned to receive one of several variant vaccines. Enrollment will target a goal of approximately 45% of each of the variant vaccine arms to be in older adults (= 65 years of age) for stages 1, 2 and 3 and approximately 20% to have had confirmed COVID-19 for all 4 stages. The primary objective is to evaluate humoral immune responses of candidate SARS-CoV-2 variant vaccines, alone or in combination.

DETAILED DESCRIPTION:
This phase 2 clinical trial will evaluate the safety and immunogenicity of additional doses of prototype and variant (alone or in combination) vaccine candidates in previously vaccinated participants with or without prior severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and will evaluate innate, cellular, and humoral immune responses to inform on how to shift the immune response to cover new variants as they emerge. A randomized open-label, non-placebo controlled, multi-site, multi-stage clinical trial in individuals, 18 years of age and older, who are in a stable state of health, has received a complete authorized/approved vaccine series (primary series + booster either with homologous or heterologous vaccine products) >/= 16 weeks prior to enrollment. Subjects will be stratified by i) age (18-64 years and = 65 years of age) (however arms 16 and 17 or stage 4 will only enroll participants between the ages of 18-49 years) and ii) history of confirmed prior SARS-CoV-2 infection, and randomly assigned to receive one of several variant vaccines. Enrollment will target a goal of approximately 45% of each of the variant vaccine arms to be in older adults (= 65 years of age) for stages 1, 2 and 3 and approximately 20% to have had confirmed COVID-19 for all 4 stages. This is an adaptive design and may add arms of new vaccine platforms and/or variant lineage spike vaccines as needed. The study arms will be conducted in different stages (that could overlap) depending on public health needs and the availability of study products (starting with the available mRNA vaccines). The primary objective is to evaluate humoral immune responses of candidate SARS-CoV-2 variant vaccines, alone or in combination. The secondary objective is to evaluate the safety of candidate SARS-CoV-2 variant vaccines, as assessed by: a) Local and systemic solicited Adverse Events for 7 days following each vaccine dose; b) Unsolicited Adverse Events from Dose 1 to 28 days following each vaccine dose; c) Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interests (AESIs), New Onset of Chronic Medical (NOCMCs) and Adverse Events (AEs) leading to withdrawal from the study from Dose 1 to 12 months after last vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible to participate in this study:

1. Individuals > / = 18 years of age at the time of consent. (18-49 years for stage 4).
2. Confirmed receipt of a complete primary and booster COVID-19 vaccine series, either homologous or heterologous, with an FDA authorized/approved vaccine at least 16 weeks prior to study vaccine dose 1.
3. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other study procedures.
4. Determined by medical history, targeted physical examination and clinical judgement of the investigator to be in stable state of health.

Note: Participants with pre-existing stable chronic medical conditions defined as condition not requiring significant change in therapy or hospitalization for worsening disease within 4 weeks from enrollment, can be included at the discretion of the investigator.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Confirmed SARS-CoV-2 infection < 16 weeks prior to any study vaccine dose.
2. Pregnant and breastfeeding participants.
3. Prior administration of an investigational coronavirus vaccine at any time or SARS-CoV-2 immunoglobulin, monoclonal antibody or plasma antibody therapy in the preceding 3 months.

   Note: subjects that participated in clinical trials of products that are now FDA approved/authorized are allowed to participate.
4. Current/planned simultaneous participation in another interventional study or receipt of any investigational study product within 28 days prior to vaccine study dose(s).
5. A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine, polyethylene glycol (PEG), polysorbate or nanolipid particles.
6. A history of myocarditis or pericarditis at any time prior to enrollment (for subjects in stages 1, 2 and 4).
7. Received or plans to receive a vaccine within 28 days prior to or after any dose of study vaccine.

   Note: Receipt of seasonal influenza vaccine is allowed at any time.
8. Bleeding disorder diagnosed by a healthcare provider (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or bleeding difficulties with intramuscular injections or blood draws.
9. Current or previous diagnosis of an immunocompromising condition or other immunosuppressive condition.
10. Advanced liver or kidney diseases.
11. Advanced (CD4 count < 200) and/or untreated HIV, untreated Hepatitis B or untreated Hepatitis C.
12. Received oral, intramuscular or intravenous systemic immunosuppressants, or immune-modifying drugs for >14 days in total within 6 months prior to any study vaccine dose (for corticosteroids = 20 mg > / = day of prednisone equivalent).

    Note: Topical medications are allowed.
13. Received immunoglobulin or blood-derived products, within 3 months prior any study vaccine dose.
14. Received chemotherapy, immunotherapy or radiation therapy within 6 months prior to any study vaccine dose.
15. Study personnel or an immediate family member or household member of study personnel.
16. Is acutely ill or febrile 72 hours prior to or at vaccine dosing (fever defined as > / = 38.0 degrees Celsius/100.4 degrees Fahrenheit). Participants meeting this criterion may be rescheduled within the relevant window periods.

    Note: Afebrile participants with minor illnesses can be enrolled at the discretion of the Investigator, as long as the illness is not suggestive of COVID-19.
17. Plan to receive a COVID-19 booster vaccine outside of the study within the next 180 days. (for subjects in Stage 4 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Alabama at Birmingham School of Medicine - Alabama Vaccine Research Clinic, Birmingham, Alabama
  - University of California, San Diego (UCSD) - Antiviral Research Center (AVRC), San Diego, California
  - Zuckerberg San Francisco General Hospital, UCSF Positive Health Program, San Francisco, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Howard University - Department of Medicine - Division of Infectious Disease, Washington D.C., District of Columbia
  - Morehouse School of Medicine - Clinical Research Center, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - The Hope Clinic of Emory University, Decatur, Georgia
  - University of Illinois at Chicago College of Medicine - Division of Infectious Diseases, Chicago, Illinois
  - University of Iowa Hospitals & Clinics - Department of Internal Medicine, Iowa City, Iowa
  - Tulane University Clinical Translational Unit, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Washington University School of Medicine in St. Louis - Infectious Disease Clinical Research Unit, St Louis, Missouri
  - NYU Grossman School, NYU Langone Vaccine Center, Long Island, Mineola, New York
  - NYU Langone Vaccine Center Research Clinic, Manhattan, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Medical Branch, League City, Texas
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Diemert DJ, Graciaa DS, Zhang B, Rouphael NG, Branche AR, Martin TCS, Jackson LA, Presti RM, Kamidani S, Mahgoub SM, Babu TM, Magaret CA, Simon V, van Bakel H, Roberts PC, Beigel JH, Gilbert PB, Follmann D; Coronavirus Variant Immunologic Landscape Trial (COVAIL) Study Team. Effect of Omicron BA.1-based compared to prototype booster mRNA vaccination on incidence of COVID-19 in the COVAIL trial. Vaccine. 2025 Oct 3;64:127718. doi: 10.1016/j.vaccine.2025.127718. Epub 2025 Sep 9. PMID 40930044
- [Derived] Fong Y, Dang L, Zhang B, Fintzi J, Chen S, Wang J, Rouphael NG, Branche AR, Diemert DJ, Falsey AR, Losada C, Baden LR, Frey SE, Whitaker JA, Little SJ, Kamidani S, Walter EB, Novak RM, Rupp R, Jackson LA, Yu C, Magaret CA, Molitor C, Borate B, Babu TM, Kottkamp AC, Luetkemeyer AF, Immergluck LC, Presti RM, Backer M, Winokur PL, Mahgoub SM, Goepfert PA, Fusco DN, Atmar RL, Posavad CM, Mu J, Makowski M, Makhene MK, Nayak SU, Roberts PC, Follmann D, Gilbert PB; Coronavirus Variant Immunologic Landscape Trial (COVAIL) Study Team. Neutralizing Antibody Immune Correlates for a Recombinant Protein Vaccine in the COVAIL Trial. Clin Infect Dis. 2025 Feb 5;80(1):223-227. doi: 10.1093/cid/ciae465. PMID 39325506
- [Derived] Branche AR, Rouphael NG, Diemert DJ, Falsey AR, Losada C, Baden LR, Frey SE, Whitaker JA, Little SJ, Anderson EJ, Walter EB, Novak RM, Rupp R, Jackson LA, Babu TM, Kottkamp AC, Luetkemeyer AF, Immergluck LC, Presti RM, Backer M, Winokur PL, Mahgoub SM, Goepfert PA, Fusco DN, Malkin E, Bethony JM, Walsh EE, Graciaa DS, Samaha H, Sherman AC, Walsh SR, Abate G, Oikonomopoulou Z, El Sahly HM, Martin TCS, Kamidani S, Smith MJ, Ladner BG, Porterfield L, Dunstan M, Wald A, Davis T, Atmar RL, Mulligan MJ, Lyke KE, Posavad CM, Meagher MA, Stephens DS, Neuzil KM, Abebe K, Hill H, Albert J, Telu K, Mu J, Lewis TC, Giebeig LA, Eaton A, Netzl A, Wilks SH, Tureli S, Makhene M, Crandon S, Montefiori DC, Makowski M, Smith DJ, Nayak SU, Roberts PC, Beigel JH; COVAIL Study Group. Comparison of bivalent and monovalent SARS-CoV-2 variant vaccines: the phase 2 randomized open-label COVAIL trial. Nat Med. 2023 Sep;29(9):2334-2346. doi: 10.1038/s41591-023-02503-4. Epub 2023 Aug 28. PMID 37640860
- [Derived] Branche A, Rouphael N, Diemert D, Falsey A, Losada C, Baden LR, Frey S, Whitaker J, Little S, Anderson E, Walter E, Novak R, Rupp R, Jackson L, Babu T, Kottkamp A, Luetkemeyer A, Immergluck L, Presti R, Backer M, Winokur P, Mahgoub S, Goepfert P, Fusco D, Malkin E, Bethony J, Walsh E, Graciaa D, Samaha H, Sherman A, Walsh S, Abate G, Oikonomopoulou Z, El Sahly H, Martin T, Kamidani S, Smith M, Ladner B, Porterfield L, Dunstan M, Wald A, Davis T, Atmar R, Mulligan M, Lyke K, Posavad C, Meagher M, Stephens D, Neuzil K, Abebe K, Hill H, Albert J, Telu K, Mu J, Lewis T, Giebeig L, Eaton A, Netzl A, Wilks S, Tureli S, Makhene M, Crandon S, Montefiori D, Makowski M, Smith D, Nayak S, Roberts P, Beigel J. Bivalent and Monovalent SARS-CoV-2 Variant Vaccine Boosters Improve coverage of the known Antigenic Landscape: Results of the COVID-19 Variant Immunologic Landscape (COVAIL) Trial. Res Sq [Preprint]. 2023 May 5:rs.3.rs-2653179. doi: 10.21203/rs.3.rs-2653179/v1. PMID 37205592
- [Derived] Branche AR, Rouphael NG, Diemert DJ, Falsey AR, Losada C, Baden LR, Frey SE, Whitaker JA, Little SJ, Anderson EJ, Walter EB, Novak RM, Rupp R, Jackson LA, Babu TM, Kottkamp AC, Luetkemeyer AF, Immergluck LC, Presti RM, Backer M, Winokur PL, Mahgoub SM, Goepfert PA, Fusco DN, Malkin E, Bethony JM, Walsh EE, Graciaa DS, Samaha H, Sherman AC, Walsh SR, Abate G, Oikonomopoulou Z, El Sahly HM, Martin TCS, Rostad CA, Smith MJ, Ladner BG, Porterfield L, Dunstan M, Wald A, Davis T, Atmar RL, Mulligan MJ, Lyke KE, Posavad CM, Meagher MA, Stephens DS, Neuzil KM, Abebe K, Hill H, Albert J, Lewis TC, Giebeig LA, Eaton A, Netzl A, Wilks SH, Tureli S, Makhene M, Crandon S, Lee M, Nayak SU, Montefiori DC, Makowski M, Smith DJ, Roberts PC, Beigel JH; COVAIL Study Group. SARS-CoV-2 Variant Vaccine Boosters Trial: Preliminary Analyses. medRxiv [Preprint]. 2022 Jul 15:2022.07.12.22277336. doi: 10.1101/2022.07.12.22277336. PMID 35898343

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 - Arm 01 (Moderna mRNA1273 Prototype): mRNA-1273 administered through 0.2 mg/ml intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike (S) protein of the B.1.351 variant SARS-CoV-2 strain.
  mRNA-1273.529: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike (S) protein of the B.1.351 variant SARS-CoV-2 strain.
  mRNA-1273.529: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron): 0.2 mg/ml of mRNA-1273.617.2 and 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273.529: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  mRNA-1273.617.2: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.617.2 (Delta) variant SARS-CoV-2 strain.
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 1 - Arm 05 (Moderna mRNA1273 Omicron): 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273.529: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype): 0.2 mg/ml of mRNA-1273.529 and mRNA-1273 0.2 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=100
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
  mRNA-1273.529: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  Sodium Chloride, 0.9%: 0.9% Sodium Chloride Injection
- Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2.
- Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2 (B.1.1.529): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
  BNT162b2 (B.1.351): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.
- Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron): 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2 (B.1.1.529): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
- Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta): 500 mcg/mL of BNT162b2 (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2 (B.1.351): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.
- Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2.
  BNT162b2 (B.1.351): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.
- Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Omicron) and 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2.
  BNT162b2 (B.1.1.529): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.
- Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype): 500 mcg/mL CoV2 preS dTM-AS03 [D614] (prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  AS03: AS03 oil-in-water emulsion adjuvant.
  CoV2 preS dTM/D614: Is a liquid formulation made of recombinant protein placed in a formulation buffer. The antigen solution contains the spike protein sequence of the ancestral strain of SARS-CoV-2.
- Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta): 500 mcg/mL CoV2 preS dTM-AS03 [B.1.351] (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  AS03: AS03 oil-in-water emulsion adjuvant.
  CoV2 preS dTM [B.1.351]: Is a liquid formulation made of recombinant protein placed in a formulation buffer that contains the spike protein sequence of the B.1.351 (Beta) variant SARS-CoV-2 strain.
- Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype): 500 mcg/mL CoV2 preS dTM-AS03 [D614 + B.1.351] (prototype + Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years) N=50
  AS03: AS03 oil-in-water emulsion adjuvant.
  CoV2 preS dTM/D614+B.1.351: Is a liquid formulation made of recombinant protein placed in a formulation buffer contains the spike protein sequences of the ancestral and B.1.351 (Beta) variant SARS-CoV-2 strains
- Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.1) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years; N=100
  BNT162b2 bivalent (wildtype and Omicron BA.1): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer. Contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.1 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2.
- Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype]): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years; N=100
  BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5): A preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer. Contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2.
Period: Overall Study
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Started | 99 | 100 | 102 | 101 | 100 | 100 | 51 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 53 | 101 | 101
Completed | 91 | 93 | 95 | 95 | 95 | 91 | 45 | 49 | 50 | 48 | 48 | 49 | 46 | 42 | 47 | 91 | 94
Not Completed | 8 | 7 | 7 | 6 | 5 | 9 | 6 | 3 | 4 | 3 | 4 | 4 | 3 | 9 | 6 | 10 | 7
Not completed — Withdrawal by Subject | 7 | 0 | 3 | 3 | 1 | 5 | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 2 | 0 | 3 | 3
Not completed — Lost to Follow-up | 1 | 4 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 4 | 2 | 7 | 4 | 6 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did not receive vaccine | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unable to make last visit | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants in Stage 1 - Arm 04 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) who did not receive second dose were analyzed as part of Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose). Participants who did not receive any vaccine were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype]) | Total
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101 | 1263
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (16.4) | 51.8 (16.9) | 53 (16.3) | 51.7 (17.5) | 52.2 (17.5) | 50.7 (18.) | 50.8 (17.6) | 50.3 (18.1) | 48.7 (16.4) | 49.9 (16.1) | 48 (17.9) | 51.7 (16) | 42.9 (18.5) | 48.7 (15.6) | 46.5 (14.7) | 31.7 (8.1) | 32.2 (8.8) | 47.6 (17.4)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 64 | 75 | 54 | 65 | 64 | 65 | 35 | 36 | 38 | 36 | 35 | 38 | 39 | 40 | 43 | 101 | 101 | 929
  >=65 years | 35 | 38 | 32 | 36 | 35 | 34 | 15 | 16 | 16 | 15 | 17 | 15 | 10 | 11 | 9 | 0 | 0 | 334
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 65 | 48 | 52 | 53 | 49 | 24 | 27 | 30 | 28 | 28 | 31 | 33 | 30 | 27 | 56 | 58 | 689
  Male | 49 | 48 | 38 | 49 | 46 | 50 | 26 | 25 | 24 | 23 | 24 | 22 | 16 | 21 | 25 | 45 | 43 | 574
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 1 | 7 | 7 | 5 | 4 | 6 | 9 | 2 | 3 | 1 | 8 | 5 | 4 | 17 | 21 | 116
  Not Hispanic or Latino | 94 | 102 | 85 | 94 | 92 | 94 | 45 | 46 | 45 | 49 | 49 | 52 | 41 | 46 | 48 | 84 | 80 | 1146
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 6
  Asian | 5 | 8 | 6 | 6 | 7 | 9 | 5 | 9 | 9 | 5 | 6 | 6 | 9 | 4 | 4 | 11 | 16 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 12 | 6 | 6 | 6 | 4 | 10 | 5 | 2 | 3 | 5 | 5 | 2 | 3 | 9 | 4 | 10 | 12 | 104
  White | 79 | 94 | 74 | 81 | 85 | 78 | 38 | 39 | 39 | 39 | 38 | 44 | 35 | 38 | 37 | 68 | 65 | 971
  More than one race | 2 | 2 | 0 | 8 | 2 | 1 | 1 | 2 | 3 | 2 | 3 | 1 | 0 | 0 | 6 | 7 | 4 | 44
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 2 | 12
Prior Infection (Self-Report) [Count of Participants; unit: Participants]
  Yes | 15 | 20 | 9 | 15 | 15 | 15 | 11 | 12 | 13 | 12 | 12 | 13 | 15 | 15 | 16 | 59 | 60 | 327
  No | 84 | 93 | 77 | 86 | 84 | 84 | 39 | 40 | 41 | 39 | 40 | 40 | 34 | 36 | 36 | 42 | 41 | 936
Prior Infection (Positive Nuclear Protein Antibody or Self-Report) [Count of Participants; unit: Participants]
  Yes | 21 | 23 | 15 | 17 | 23 | 20 | 17 | 18 | 18 | 18 | 15 | 18 | 22 | 20 | 20 | 80 | 76 | 441
  No | 78 | 90 | 71 | 84 | 76 | 79 | 33 | 34 | 36 | 33 | 37 | 35 | 27 | 31 | 32 | 21 | 25 | 822
SARS-COV-2 Vaccination Regimen [Count of Participants; unit: Participants]
  mRNA Primary, mRNA Boost | 95 | 107 | 82 | 95 | 95 | 96 | 50 | 52 | 54 | 50 | 52 | 51 | 46 | 50 | 50 | 94 | 94 | 1213
  Ad26 Primary, mRNA Boost | 4 | 6 | 3 | 5 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 6 | 6 | 42
  Ad26 Primary, Ad26 Boost | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 8
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.69 (5.41) | 27.38 (5.95) | 27.17 (5.4) | 27.27 (5.41) | 27.17 (5.69) | 27.14 (5.46) | 26.38 (3.51) | 28.17 (6.45) | 26.81 (6.78) | 28.42 (6.11) | 27.54 (6.33) | 28.88 (5.98) | 25.87 (5.91) | 28.85 (6.7) | 27.77 (6.35) | 26.95 (5.58) | 27.18 (6.15) | 27.47 (5.83)
Days Since Most Recent COVID19 Vaccine [Mean (Standard Deviation); unit: days] | 172.8 (32.3) | 165.5 (27.7) | 175.5 (23.8) | 170.3 (29.3) | 173.2 (28.1) | 168.6 (27.2) | 195.5 (33.6) | 196.6 (34.2) | 200.2 (35.6) | 207.5 (31.7) | 207.2 (29.3) | 198.3 (34.6) | 205.9 (38.1) | 194.3 (40.9) | 210.9 (41.2) | 332.5 (44.5) | 334 (66.1) | 208.2 (67.3)
Days Since Most Recent Self-Reported COVID19 Infection [Mean (Standard Deviation); unit: days] | 389.1 (236) | 327.7 (206.1) | 358.7 (246.8) | 329.4 (214.2) | 425.9 (243.3) | 334.1 (198.4) | 240.8 (174.1) | 373.1 (280.1) | 242.8 (139.4) | 250.8 (163.8) | 314.2 (251.1) | 219.2 (192) | 224.7 (174.4) | 224.4 (93.4) | 275.1 (235.5) | 292.1 (197.1) | 304.5 (191.7) | 301.3 (204.3)
Days Since Most Recent Self-Reported COVID19 Infection or COVID19 Vaccine [Mean (Standard Deviation); unit: days] | 169.2 (33.8) | 162.5 (28.1) | 173.5 (25.8) | 167.8 (30.3) | 170.8 (30) | 166.7 (27.6) | 190.5 (37.3) | 189.2 (38.5) | 193.4 (40) | 198.3 (38.3) | 196.8 (38.1) | 188.9 (40.5) | 195.1 (44.1) | 183.4 (40.5) | 195.4 (47.9) | 269.8 (82.3) | 274 (83.2) | 193.6 (58.2)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against Wa-1 in One Dose Groups.
Description: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against Wa-1. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 29, Day 91, Day 181, Day 271, Day 366
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported. Participants in Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) who did not receive second dose were analyzed as part of Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose).
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- Stage 1 - Arm 01 (Moderna mRNA1273 Prototype): mRNA-1273 administered through 0.2 mg/ml intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron): 0.2 mg/ml of mRNA-1273.617.2 and 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 1 - Arm 05 (Moderna mRNA1273 Omicron): 0.2 mg/ml of mRNA-1273.529 administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype): 0.2 mg/ml of mRNA-1273.529 and mRNA-1273 0.2 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron): 500 mcg/mL of BNT162b2 (Omicron) administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta): 500 mcg/mL of BNT162b2 (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Beta) and 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]): 500 mcg/mL of BNT162b2 (Omicron) and 500 mcg/mL of BNT162b2 (Wildtype [Prototype]) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype): 500 mcg/mL CoV2 preS dTM-AS03 [D614] (prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta): 500 mcg/mL CoV2 preS dTM-AS03 [B.1.351] (Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype): 500 mcg/mL CoV2 preS dTM-AS03 [D614 + B.1.351] (prototype + Beta) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
- Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.1) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years;
- Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype]): 100 mcg/mL BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5) + Wildtype (Prototype) administered through intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 49 years;
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 98 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 29: number analyzed (Participants) | 88 | 110 | 96 | 94 | 86 | 45 | 51 | 47 | 50 | 50 | 45 | 45 | 43 | 50 | 95 | 95
  Day 29 | 4.57 [3.85 to 5.43] | 3.61 [3.17 to 4.11] | 3.78 [3.24 to 4.40] | 3.87 [3.32 to 4.51] | 3.67 [3.15 to 4.28] | 3.25 [2.64 to 4.00] | 3.75 [3.15 to 4.45] | 3.55 [2.82 to 4.46] | 4.25 [3.55 to 5.10] | 4.09 [3.39 to 4.93] | 4.19 [3.41 to 5.15] | 2.24 [1.88 to 2.67] | 2.59 [2.06 to 3.25] | 2.30 [1.87 to 2.84] | 3.05 [2.65 to 3.50] | 3.29 [2.87 to 3.77]
  Day 91: number analyzed (Participants) | 91 | 108 | 94 | 93 | 91 | 47 | 49 | 48 | 47 | 46 | 48 | 45 | 45 | 50 | 97 | 96
  Day 91 | 2.59 [2.18 to 3.08] | 2.42 [2.13 to 2.75] | 2.65 [2.24 to 3.13] | 2.74 [2.34 to 3.21] | 2.55 [2.17 to 3.00] | 2.44 [1.88 to 3.18] | 2.62 [2.16 to 3.16] | 2.43 [1.97 to 3.00] | 3.03 [2.47 to 3.71] | 2.64 [2.21 to 3.15] | 2.61 [2.14 to 3.19] | 1.72 [1.33 to 2.23] | 2.22 [1.70 to 2.91] | 1.93 [1.49 to 2.50] | 2.03 [1.77 to 2.34] | 2.28 [2.01 to 2.58]
  Day 181: number analyzed (Participants) | 91 | 105 | 95 | 96 | 92 | 41 | 49 | 46 | 48 | 49 | 44 | 44 | 40 | 48 | 94 | 95
  Day 181 | 1.85 [1.51 to 2.28] | 1.75 [1.48 to 2.07] | 1.73 [1.42 to 2.10] | 1.86 [1.55 to 2.22] | 1.90 [1.57 to 2.28] | 2.04 [1.44 to 2.88] | 1.68 [1.34 to 2.10] | 1.65 [1.26 to 2.17] | 2.16 [1.63 to 2.85] | 1.93 [1.54 to 2.41] | 1.47 [1.13 to 1.92] | 1.71 [1.28 to 2.28] | 1.95 [1.47 to 2.58] | 1.89 [1.38 to 2.57] | 1.46 [1.26 to 1.69] | 1.68 [1.44 to 1.97]
  Day 271: number analyzed (Participants) | 90 | 96 | 90 | 95 | 87 | 40 | 49 | 48 | 46 | 47 | 48 | 44 | 42 | 45 | 87 | 94
  Day 271 | 2.41 [1.93 to 3.00] | 2.05 [1.70 to 2.48] | 2.19 [1.78 to 2.69] | 2.41 [1.95 to 2.97] | 2.18 [1.78 to 2.67] | 2.23 [1.57 to 3.18] | 1.97 [1.56 to 2.50] | 1.72 [1.28 to 2.30] | 2.60 [1.91 to 3.54] | 2.16 [1.66 to 2.82] | 1.81 [1.36 to 2.41] | 1.92 [1.38 to 2.67] | 2.05 [1.54 to 2.73] | 1.75 [1.27 to 2.40] | 1.20 [1.02 to 1.41] | 1.25 [1.06 to 1.47]
  Day 366: number analyzed (Participants) | 85 | 96 | 93 | 91 | 89 | 42 | 48 | 48 | 45 | 45 | 44 | 45 | 40 | 45 | 89 | 90
  Day 366 | 2.01 [1.65 to 2.46] | 1.88 [1.55 to 2.28] | 1.85 [1.50 to 2.29] | 1.78 [1.45 to 2.19] | 1.61 [1.32 to 1.96] | 1.43 [1.03 to 1.98] | 1.52 [1.17 to 1.97] | 1.26 [0.96 to 1.66] | 1.74 [1.28 to 2.38] | 1.72 [1.32 to 2.25] | 1.50 [1.10 to 2.05] | 1.31 [0.92 to 1.87] | 1.41 [1.07 to 1.86] | 1.28 [0.92 to 1.78] | 1.06 [0.89 to 1.25] | 1.08 [0.93 to 1.26]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against Wa-1 in Two Dose Group.
Description: as for outcome 1
Time Frame: Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses): 0.1 mg/ml of mRNA-1273.351 and 0.2 mg/ml of mRNA-1273.529 mg/ml administered through intramuscular injection in the deltoid muscle on Day 1 and Day 57 in participants from 18 to 64; > / = 65 years (~45% in > / = 65 years)
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 29: number analyzed (Participants) | 77
  Day 29 | 4.09 [3.48 to 4.81]
  Day 57: number analyzed (Participants) | 79
  Day 57 | 3.02 [2.59 to 3.52]
  Day 85: number analyzed (Participants) | 77
  Day 85 | 4.85 [4.09 to 5.75]
  Day 147: number analyzed (Participants) | 78
  Day 147 | 3.74 [3.11 to 4.51]
  Day 237: number analyzed (Participants) | 82
  Day 237 | 2.68 [2.16 to 3.32]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2.31 [1.84 to 2.89]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 1.75 [1.37 to 2.23]

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against B.1.351 in One Dose Groups.
Description: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against B.1.351. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 29: number analyzed (Participants) | 96 | 110 | 94 | 93 | 91 | 48 | 49 | 49 | 50 | 47 | 46 | 46 | 44 | 50 | 98 | 95
  Day 29 | 4.66 [3.93 to 5.51] | 4.31 [3.71 to 4.99] | 4.50 [3.84 to 5.29] | 4.96 [4.22 to 5.83] | 4.28 [3.58 to 5.12] | 3.59 [2.95 to 4.37] | 5.31 [4.39 to 6.41] | 4.35 [3.39 to 5.57] | 5.58 [4.63 to 6.73] | 5.25 [4.34 to 6.35] | 5.01 [4.02 to 6.25] | 2.31 [1.92 to 2.79] | 3.07 [2.42 to 3.89] | 2.68 [2.13 to 3.38] | 3.59 [3.17 to 4.07] | 3.75 [3.22 to 4.38]
  Day 91: number analyzed (Participants) | 91 | 110 | 96 | 97 | 94 | 48 | 50 | 49 | 48 | 49 | 49 | 47 | 47 | 51 | 98 | 97
  Day 91 | 2.81 [2.33 to 3.39] | 2.85 [2.49 to 3.26] | 2.99 [2.51 to 3.56] | 3.28 [2.80 to 3.85] | 3.00 [2.52 to 3.57] | 2.58 [2.00 to 3.32] | 3.31 [2.75 to 3.99] | 2.85 [2.29 to 3.55] | 3.76 [3.09 to 4.57] | 3.48 [2.79 to 4.33] | 3.06 [2.41 to 3.87] | 1.77 [1.34 to 2.33] | 2.50 [1.93 to 3.24] | 2.12 [1.60 to 2.81] | 2.23 [1.96 to 2.54] | 2.55 [2.20 to 2.96]
  Day 181: number analyzed (Participants) | 91 | 105 | 97 | 96 | 94 | 41 | 49 | 47 | 50 | 50 | 45 | 44 | 41 | 49 | 94 | 94
  Day 181 | 1.87 [1.52 to 2.30] | 1.90 [1.62 to 2.24] | 1.92 [1.56 to 2.35] | 2.05 [1.72 to 2.45] | 2.04 [1.69 to 2.47] | 2.19 [1.51 to 3.17] | 1.91 [1.51 to 2.42] | 1.85 [1.38 to 2.49] | 2.46 [1.86 to 3.26] | 2.06 [1.66 to 2.57] | 1.65 [1.23 to 2.22] | 1.82 [1.29 to 2.57] | 2.29 [1.73 to 3.03] | 2.15 [1.55 to 2.98] | 1.69 [1.47 to 1.95] | 1.97 [1.64 to 2.36]
  Day 271: number analyzed (Participants) | 89 | 98 | 90 | 96 | 88 | 41 | 49 | 49 | 46 | 47 | 49 | 44 | 41 | 45 | 87 | 94
  Day 271 | 2.83 [2.25 to 3.54] | 2.59 [2.12 to 3.15] | 2.79 [2.24 to 3.47] | 2.90 [2.34 to 3.59] | 2.70 [2.16 to 3.36] | 2.69 [1.88 to 3.85] | 2.42 [1.90 to 3.09] | 1.95 [1.44 to 2.65] | 3.15 [2.30 to 4.30] | 2.64 [1.97 to 3.53] | 2.23 [1.61 to 3.10] | 2.12 [1.48 to 3.04] | 2.46 [1.83 to 3.30] | 2.09 [1.49 to 2.92] | 1.35 [1.14 to 1.59] | 1.37 [1.15 to 1.64]
  Day 366: number analyzed (Participants) | 89 | 101 | 94 | 95 | 90 | 44 | 48 | 48 | 46 | 47 | 46 | 46 | 40 | 45 | 89 | 90
  Day 366 | 2.50 [2.01 to 3.11] | 2.31 [1.90 to 2.79] | 2.26 [1.81 to 2.82] | 2.18 [1.75 to 2.71] | 1.83 [1.49 to 2.25] | 1.71 [1.20 to 2.44] | 1.81 [1.36 to 2.42] | 1.34 [1.00 to 1.79] | 1.98 [1.44 to 2.72] | 2.10 [1.56 to 2.83] | 1.86 [1.33 to 2.61] | 1.48 [1.00 to 2.18] | 1.68 [1.25 to 2.27] | 1.45 [1.03 to 2.04] | 1.16 [0.97 to 1.38] | 1.16 [0.97 to 1.38]

4. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against B.1.351 in Two Dose Group.
Description: as for outcome 3
Time Frame: Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 29: number analyzed (Participants) | 78
  Day 29 | 5.30 [4.49 to 6.25]
  Day 57: number analyzed (Participants) | 80
  Day 57 | 4.07 [3.48 to 4.76]
  Day 85: number analyzed (Participants) | 77
  Day 85 | 6.61 [5.48 to 7.97]
  Day 147: number analyzed (Participants) | 83
  Day 147 | 4.55 [3.78 to 5.47]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 3.44 [2.74 to 4.31]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2.91 [2.30 to 3.70]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 2.15 [1.66 to 2.77]

5. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against BA.1 in One Dose Groups.
Description: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against BA.1. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 29: number analyzed (Participants) | 97 | 112 | 99 | 98 | 93 | 48 | 51 | 50 | 50 | 51 | 52 | 46 | 46 | 51 | 99 | 98
  Day 29 | 5.24 [4.40 to 6.25] | 4.95 [4.22 to 5.81] | 5.35 [4.47 to 6.39] | 6.19 [5.30 to 7.24] | 5.30 [4.49 to 6.24] | 3.89 [3.16 to 4.79] | 6.37 [5.29 to 7.67] | 5.71 [4.47 to 7.30] | 6.20 [5.10 to 7.54] | 5.64 [4.54 to 7.01] | 6.03 [4.83 to 7.52] | 2.67 [2.19 to 3.26] | 3.36 [2.63 to 4.29] | 2.86 [2.28 to 3.59] | 4.48 [3.93 to 5.10] | 4.81 [4.06 to 5.69]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 3.06 [2.53 to 3.71] | 3.05 [2.64 to 3.52] | 3.36 [2.80 to 4.04] | 3.87 [3.27 to 4.58] | 3.38 [2.82 to 4.07] | 2.51 [1.91 to 3.30] | 3.58 [2.94 to 4.36] | 3.43 [2.72 to 4.32] | 3.93 [3.15 to 4.91] | 3.48 [2.76 to 4.39] | 3.17 [2.52 to 3.98] | 1.95 [1.44 to 2.64] | 2.32 [1.79 to 3.02] | 2.08 [1.57 to 2.76] | 2.65 [2.32 to 3.04] | 2.82 [2.42 to 3.29]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 45 | 43 | 50 | 94 | 95
  Day 181 | 1.90 [1.52 to 2.38] | 1.94 [1.63 to 2.32] | 1.93 [1.56 to 2.39] | 2.20 [1.83 to 2.65] | 2.17 [1.77 to 2.65] | 2.24 [1.53 to 3.28] | 2.18 [1.72 to 2.78] | 2.22 [1.66 to 2.95] | 2.44 [1.86 to 3.21] | 2.04 [1.60 to 2.61] | 1.90 [1.37 to 2.63] | 1.88 [1.32 to 2.69] | 2.30 [1.73 to 3.06] | 2.03 [1.47 to 2.80] | 1.87 [1.61 to 2.17] | 2.05 [1.70 to 2.47]
  Day 271: number analyzed (Participants) | 90 | 100 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 45 | 43 | 47 | 87 | 94
  Day 271 | 2.80 [2.21 to 3.56] | 2.64 [2.14 to 3.26] | 2.95 [2.31 to 3.77] | 3.17 [2.52 to 3.98] | 2.90 [2.30 to 3.66] | 2.52 [1.75 to 3.62] | 2.65 [2.05 to 3.43] | 2.25 [1.66 to 3.07] | 3.15 [2.31 to 4.29] | 2.65 [1.96 to 3.59] | 2.31 [1.66 to 3.21] | 2.30 [1.58 to 3.35] | 2.40 [1.78 to 3.23] | 2.06 [1.47 to 2.88] | 1.37 [1.14 to 1.64] | 1.32 [1.10 to 1.59]
  Day 366: number analyzed (Participants) | 89 | 100 | 95 | 95 | 90 | 44 | 48 | 49 | 48 | 47 | 47 | 46 | 39 | 45 | 89 | 90
  Day 366 | 2.33 [1.85 to 2.94] | 2.24 [1.81 to 2.77] | 2.27 [1.79 to 2.88] | 2.29 [1.81 to 2.91] | 1.87 [1.49 to 2.34] | 1.55 [1.09 to 2.19] | 1.90 [1.41 to 2.55] | 1.55 [1.11 to 2.17] | 2.14 [1.50 to 3.06] | 2.07 [1.52 to 2.81] | 1.95 [1.36 to 2.80] | 1.38 [0.91 to 2.09] | 1.46 [1.07 to 1.99] | 1.36 [0.95 to 1.94] | 1.19 [0.99 to 1.44] | 1.13 [0.94 to 1.37]

6. Primary Outcome: Geometric Mean Fold Rise (GMFR) of AUC From Baseline Antibody Against BA.1 in Two Dose Group.
Description: as for outcome 5
Time Frame: Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 29: number analyzed (Participants) | 85
  Day 29 | 5.96 [4.99 to 7.11]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 4.69 [3.94 to 5.59]
  Day 85: number analyzed (Participants) | 83
  Day 85 | 7.99 [6.54 to 9.76]
  Day 147 | 5.28 [4.30 to 6.49]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 3.47 [2.71 to 4.43]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2.91 [2.24 to 3.77]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 2.03 [1.54 to 2.68]

7. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against D614G in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against D614G. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 6.49 [5.40 to 7.81] | 5.41 [4.38 to 6.68] | 6.88 [5.29 to 8.94] | 4.98 [4.00 to 6.21] | 7.31 [5.64 to 9.47] | 4.27 [3.26 to 5.58] | 3.99 [3.15 to 5.07] | 3.98 [3.07 to 5.17] | 5.11 [3.94 to 6.63] | 4.89 [3.94 to 6.07] | 6.12 [4.34 to 8.62] | 1.57 [1.28 to 1.92] | 2.82 [1.72 to 4.63] | 1.84 [1.41 to 2.40] | 3.69 [3.10 to 4.39] | 4.33 [3.49 to 5.37]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 4.80 [3.97 to 5.80] | 4.25 [3.44 to 5.24] | 5.07 [3.87 to 6.64] | 3.77 [3.05 to 4.68] | 4.97 [3.92 to 6.29] | 3.45 [2.60 to 4.58] | 4.25 [3.09 to 5.86] | 3.85 [3.03 to 4.89] | 4.25 [3.16 to 5.72] | 4.46 [3.52 to 5.64] | 5.09 [3.63 to 7.14] | 2.00 [1.62 to 2.46] | 4.26 [2.46 to 7.36] | 2.72 [2.02 to 3.65] | 4.20 [3.55 to 4.97] | 4.64 [3.73 to 5.78]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 3.50 [2.67 to 4.58] | 3.74 [3.03 to 4.60] | 4.45 [3.46 to 5.72] | 3.70 [2.92 to 4.67] | 4.71 [3.53 to 6.29] | 1.92 [1.32 to 2.79] | 2.03 [1.51 to 2.72] | 2.11 [1.60 to 2.78] | 2.29 [1.67 to 3.13] | 2.19 [1.67 to 2.88] | 2.48 [1.73 to 3.56] | 2.21 [1.59 to 3.06] | 3.75 [2.08 to 6.76] | 2.20 [1.53 to 3.17] | 1.93 [1.64 to 2.27] | 2.46 [2.01 to 3.02]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 2.05 [1.52 to 2.76] | 2.00 [1.56 to 2.56] | 2.52 [1.88 to 3.39] | 1.97 [1.54 to 2.52] | 2.85 [2.10 to 3.87] | 2.61 [1.60 to 4.27] | 1.82 [1.28 to 2.58] | 1.82 [1.26 to 2.64] | 2.18 [1.47 to 3.24] | 1.99 [1.48 to 2.68] | 2.23 [1.43 to 3.49] | 2.36 [1.59 to 3.51] | 3.02 [1.75 to 5.21] | 2.48 [1.68 to 3.67] | 1.46 [1.20 to 1.78] | 1.57 [1.27 to 1.94]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 3.44 [2.50 to 4.73] | 3.41 [2.52 to 4.61] | 3.54 [2.60 to 4.82] | 3.09 [2.34 to 4.07] | 3.59 [2.66 to 4.86] | 2.82 [1.74 to 4.57] | 2.24 [1.62 to 3.10] | 1.86 [1.31 to 2.65] | 3.10 [2.00 to 4.82] | 2.21 [1.45 to 3.37] | 2.39 [1.70 to 3.36] | 2.43 [1.58 to 3.73] | 3.44 [1.86 to 6.36] | 2.30 [1.52 to 3.49] | 1.23 [0.99 to 1.52] | 1.33 [1.09 to 1.63]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 2.77 [2.11 to 3.63] | 2.29 [1.75 to 3.00] | 2.44 [1.85 to 3.20] | 2.09 [1.60 to 2.74] | 2.60 [1.90 to 3.55] | 2.59 [1.64 to 4.09] | 2.20 [1.53 to 3.18] | 1.73 [1.15 to 2.59] | 2.76 [1.77 to 4.29] | 2.88 [2.03 to 4.09] | 3.08 [1.96 to 4.83] | 2.43 [1.60 to 3.69] | 3.65 [1.90 to 7.00] | 2.43 [1.65 to 3.60] | 1.08 [0.87 to 1.35] | 1.13 [0.92 to 1.39]

8. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against D614G in Two Dose Group.
Description: as for outcome 7
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 15 | 5.35 [4.45 to 6.43]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 3.81 [2.93 to 4.95]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 3.33 [2.78 to 3.99]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 4.88 [3.99 to 5.97]
  Day 147 | 2.97 [2.35 to 3.76]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 3.73 [2.77 to 5.02]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2.67 [1.98 to 3.60]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 3.02 [2.19 to 4.16]

9. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against B.1.351 in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against B.1.351. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported. Participants in Stage 1 - Arm 04 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) who did not receive second dose were analyzed as part of Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose).
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 9.47 [7.56 to 11.86] | 12.48 [10.10 to 15.41] | 11.51 [8.75 to 15.13] | 12.01 [9.39 to 15.36] | 11.23 [8.70 to 14.49] | 5.70 [4.16 to 7.83] | 8.02 [5.80 to 11.09] | 9.67 [6.77 to 13.81] | 10.69 [7.67 to 14.91] | 8.11 [6.05 to 10.86] | 10.42 [6.84 to 15.88] | 2.05 [1.47 to 2.85] | 5.91 [3.39 to 10.29] | 3.14 [2.05 to 4.82] | 5.50 [4.52 to 6.70] | 6.63 [5.22 to 8.43]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 5.69 [4.60 to 7.04] | 9.14 [7.52 to 11.11] | 7.72 [5.82 to 10.26] | 8.20 [6.50 to 10.34] | 7.15 [5.73 to 8.92] | 4.30 [3.08 to 6.01] | 7.53 [5.40 to 10.50] | 9.31 [6.57 to 13.20] | 9.22 [6.58 to 12.92] | 6.77 [4.89 to 9.39] | 8.52 [5.70 to 12.74] | 2.86 [2.09 to 3.91] | 10.37 [5.75 to 18.71] | 5.10 [3.26 to 7.98] | 4.84 [3.99 to 5.87] | 5.68 [4.45 to 7.26]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 4.31 [3.27 to 5.69] | 6.73 [5.42 to 8.35] | 6.34 [4.71 to 8.54] | 7.18 [5.53 to 9.32] | 6.96 [5.15 to 9.41] | 2.35 [1.49 to 3.70] | 3.71 [2.53 to 5.44] | 4.67 [3.26 to 6.68] | 4.65 [3.18 to 6.81] | 3.53 [2.44 to 5.10] | 4.71 [2.93 to 7.58] | 2.94 [1.83 to 4.73] | 8.23 [4.39 to 15.42] | 3.72 [2.17 to 6.38] | 2.16 [1.77 to 2.64] | 2.72 [2.16 to 3.42]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 2.41 [1.76 to 3.29] | 3.35 [2.37 to 4.74] | 3.26 [2.36 to 4.49] | 3.62 [2.63 to 4.98] | 4.36 [3.09 to 6.15] | 3.01 [1.63 to 5.58] | 2.61 [1.71 to 4.00] | 2.86 [1.79 to 4.56] | 3.25 [2.10 to 5.03] | 2.28 [1.56 to 3.33] | 3.03 [1.76 to 5.24] | 2.90 [1.65 to 5.12] | 5.31 [2.90 to 9.71] | 3.89 [2.27 to 6.67] | 1.95 [1.51 to 2.52] | 2.07 [1.60 to 2.68]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 4.15 [2.92 to 5.91] | 4.89 [3.41 to 7.00] | 4.50 [3.22 to 6.27] | 4.70 [3.44 to 6.42] | 5.11 [3.66 to 7.15] | 4.70 [2.59 to 8.55] | 4.21 [2.79 to 6.36] | 3.39 [2.21 to 5.22] | 5.09 [3.12 to 8.29] | 3.94 [2.38 to 6.52] | 5.21 [3.11 to 8.75] | 3.94 [2.21 to 7.03] | 7.86 [4.11 to 15.02] | 4.26 [2.38 to 7.63] | 1.20 [0.93 to 1.54] | 1.23 [0.96 to 1.59]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 3.62 [2.54 to 5.15] | 3.67 [2.66 to 5.06] | 3.22 [2.35 to 4.42] | 3.33 [2.35 to 4.71] | 3.50 [2.51 to 4.89] | 3.36 [1.88 to 6.01] | 3.22 [2.03 to 5.11] | 2.76 [1.73 to 4.40] | 4.10 [2.44 to 6.91] | 3.46 [2.19 to 5.48] | 4.84 [2.74 to 8.54] | 3.04 [1.75 to 5.28] | 4.79 [2.61 to 8.81] | 3.15 [1.90 to 5.22] | 1.41 [1.08 to 1.84] | 1.45 [1.11 to 1.89]

10. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against B.1.351 in Two Dose Group.
Description: as for outcome 9
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 15 | 13.31 [10.46 to 16.95]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 9.27 [7.38 to 11.64]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 7.10 [5.63 to 8.97]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 12.37 [9.48 to 16.16]
  Day 147 | 5.98 [4.45 to 8.02]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 6.60 [4.72 to 9.22]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 5.17 [3.65 to 7.31]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 4.49 [3.08 to 6.53]

11. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against B.1.617.2 in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against B.1.617.2. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 7.22 [5.89 to 8.84] | 7.26 [5.84 to 9.03] | 8.18 [6.25 to 10.69] | 6.10 [4.87 to 7.63] | 7.89 [6.15 to 10.12] | 4.50 [3.36 to 6.03] | 4.95 [3.80 to 6.44] | 4.93 [3.61 to 6.75] | 5.15 [3.93 to 6.74] | 5.15 [3.94 to 6.72] | 6.54 [4.69 to 9.13] | 1.37 [1.10 to 1.71] | 2.86 [1.75 to 4.68] | 1.93 [1.32 to 2.84] | 4.41 [3.71 to 5.23] | 5.00 [4.03 to 6.22]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 4.80 [3.91 to 5.90] | 5.29 [4.23 to 6.61] | 6.02 [4.61 to 7.88] | 4.40 [3.50 to 5.54] | 5.51 [4.31 to 7.05] | 3.73 [2.74 to 5.08] | 5.19 [3.78 to 7.12] | 4.72 [3.48 to 6.41] | 4.90 [3.67 to 6.56] | 4.82 [3.68 to 6.30] | 5.65 [4.08 to 7.83] | 2.15 [1.70 to 2.72] | 5.32 [3.08 to 9.17] | 3.55 [2.40 to 5.26] | 4.04 [3.43 to 4.77] | 4.48 [3.62 to 5.55]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 3.25 [2.44 to 4.33] | 4.46 [3.61 to 5.51] | 4.45 [3.41 to 5.80] | 3.85 [3.07 to 4.83] | 5.01 [3.76 to 6.67] | 2.22 [1.50 to 3.29] | 2.59 [1.88 to 3.56] | 2.81 [2.03 to 3.89] | 2.57 [1.84 to 3.58] | 2.34 [1.73 to 3.17] | 3.07 [2.12 to 4.46] | 2.07 [1.45 to 2.94] | 4.17 [2.33 to 7.47] | 2.59 [1.63 to 4.13] | 1.88 [1.58 to 2.25] | 2.28 [1.86 to 2.78]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 1.79 [1.33 to 2.42] | 2.03 [1.52 to 2.71] | 2.16 [1.63 to 2.85] | 1.86 [1.44 to 2.40] | 2.41 [1.83 to 3.18] | 2.23 [1.32 to 3.76] | 1.72 [1.22 to 2.44] | 1.83 [1.23 to 2.72] | 1.81 [1.21 to 2.71] | 1.71 [1.25 to 2.32] | 1.88 [1.22 to 2.88] | 1.81 [1.21 to 2.71] | 3.06 [1.75 to 5.37] | 2.54 [1.58 to 4.06] | 1.65 [1.35 to 2.02] | 1.85 [1.49 to 2.30]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 2.97 [2.14 to 4.13] | 3.07 [2.29 to 4.10] | 2.80 [2.08 to 3.76] | 2.66 [1.98 to 3.57] | 3.04 [2.24 to 4.14] | 2.72 [1.64 to 4.48] | 2.28 [1.57 to 3.31] | 1.92 [1.35 to 2.72] | 2.72 [1.73 to 4.29] | 2.17 [1.40 to 3.37] | 2.59 [1.74 to 3.85] | 2.34 [1.56 to 3.51] | 3.73 [1.99 to 7.01] | 2.53 [1.51 to 4.24] | 1.29 [1.05 to 1.59] | 1.34 [1.08 to 1.66]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 2.55 [1.90 to 3.43] | 2.45 [1.88 to 3.21] | 2.29 [1.76 to 2.96] | 1.96 [1.48 to 2.59] | 2.27 [1.67 to 3.09] | 2.45 [1.52 to 3.93] | 2.28 [1.49 to 3.48] | 1.82 [1.26 to 2.64] | 2.53 [1.60 to 3.99] | 2.59 [1.73 to 3.88] | 3.18 [1.96 to 5.16] | 1.88 [1.23 to 2.86] | 2.96 [1.68 to 5.23] | 2.44 [1.51 to 3.95] | 1.54 [1.22 to 1.95] | 1.61 [1.30 to 2.00]

12. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against B.1.617.2 in Two Dose Group.
Description: as for outcome 11
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 15 | 6.72 [5.41 to 8.35]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 4.98 [4.01 to 6.19]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 4.15 [3.30 to 5.23]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 6.60 [5.17 to 8.42]
  Day 147 | 3.32 [2.58 to 4.28]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 3.43 [2.52 to 4.66]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2.61 [1.89 to 3.60]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 2.64 [1.89 to 3.69]

13. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against BA.1 in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against BA.1. Fold-rise is calculated by dividing post-vaccination results by the baseline value The geometric mean of the fold rise is then reported
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 10.10 [7.93 to 12.85] | 16.85 [12.59 to 22.54] | 16.34 [12.20 to 21.89] | 17.50 [13.41 to 22.83] | 15.32 [11.57 to 20.29] | 5.93 [4.14 to 8.49] | 12.07 [8.50 to 17.13] | 14.51 [10.02 to 20.99] | 12.23 [8.47 to 17.65] | 9.37 [6.69 to 13.12] | 15.15 [9.61 to 23.89] | 2.98 [2.17 to 4.10] | 6.74 [4.12 to 11.03] | 4.28 [3.11 to 5.90] | 5.95 [4.86 to 7.28] | 6.49 [5.16 to 8.18]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 97 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 6.84 [5.38 to 8.69] | 12.75 [9.65 to 16.84] | 11.63 [8.59 to 15.76] | 12.07 [9.37 to 15.55] | 10.40 [8.03 to 13.47] | 3.81 [2.67 to 5.44] | 8.26 [5.82 to 11.71] | 11.70 [7.98 to 17.15] | 8.49 [6.04 to 11.92] | 7.07 [5.03 to 9.95] | 9.40 [6.04 to 14.63] | 2.59 [1.65 to 4.06] | 8.72 [4.95 to 15.36] | 4.94 [3.29 to 7.42] | 4.70 [3.90 to 5.65] | 5.10 [4.03 to 6.43]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 4.12 [3.05 to 5.56] | 8.18 [6.24 to 10.73] | 7.84 [5.80 to 10.61] | 6.94 [5.21 to 9.26] | 7.24 [5.41 to 9.70] | 3.02 [1.78 to 5.11] | 6.27 [4.07 to 9.67] | 9.44 [6.33 to 14.09] | 6.44 [4.22 to 9.83] | 5.15 [3.30 to 8.03] | 8.01 [4.86 to 13.20] | 3.02 [1.80 to 5.04] | 6.29 [3.82 to 10.35] | 3.91 [2.42 to 6.32] | 3.52 [2.86 to 4.32] | 4.02 [3.13 to 5.18]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 2.72 [1.93 to 3.83] | 5.23 [3.71 to 7.38] | 4.52 [3.17 to 6.44] | 4.84 [3.47 to 6.74] | 5.17 [3.70 to 7.23] | 4.08 [2.04 to 8.15] | 4.20 [2.36 to 7.46] | 5.32 [3.39 to 8.35] | 4.84 [3.00 to 7.81] | 3.66 [2.34 to 5.73] | 5.15 [2.89 to 9.17] | 4.58 [2.68 to 7.83] | 7.92 [4.51 to 13.90] | 6.17 [3.83 to 9.93] | 2.95 [2.28 to 3.80] | 3.23 [2.42 to 4.30]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 5.77 [4.01 to 8.28] | 8.21 [5.76 to 11.69] | 8.76 [5.96 to 12.87] | 7.40 [5.26 to 10.42] | 8.20 [5.73 to 11.75] | 6.42 [3.39 to 12.17] | 7.53 [4.89 to 11.60] | 6.14 [3.75 to 10.06] | 7.09 [4.23 to 11.88] | 5.54 [3.30 to 9.30] | 8.36 [4.74 to 14.75] | 6.35 [3.61 to 11.17] | 7.00 [3.96 to 12.38] | 6.26 [3.59 to 10.94] | 2.33 [1.79 to 3.02] | 2.33 [1.75 to 3.11]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 4.84 [3.34 to 7.02] | 7.30 [5.11 to 10.44] | 7.18 [4.92 to 10.48] | 5.94 [4.10 to 8.62] | 5.64 [3.93 to 8.10] | 4.75 [2.48 to 9.09] | 7.10 [4.32 to 11.69] | 6.36 [3.78 to 10.67] | 6.56 [3.89 to 11.08] | 6.67 [4.07 to 10.92] | 11.14 [6.02 to 20.61] | 5.13 [2.90 to 9.09] | 6.75 [4.06 to 11.20] | 5.86 [3.45 to 9.93] | 2.24 [1.69 to 2.98] | 2.09 [1.58 to 2.77]

14. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against BA.1 in Two Dose Group.
Description: Pseudovirus Neutralization From Baseline Against BA.1. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 15 | 17.18 [13.24 to 22.28]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 12.96 [9.89 to 17.00]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 9.08 [6.98 to 11.79]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 16.67 [12.55 to 22.14]
  Day 147 | 10.48 [7.92 to 13.87]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 8.78 [6.13 to 12.58]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 8.29 [5.70 to 12.06]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 8.79 [5.89 to 13.12]

15. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against BA.2.12.1 in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against BA.2.12.1. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 15
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported. Participants in Stage 1 - Arm 03 who did not receive second dose were analyzed as part of Stage 1 - Arm 02. BA.2.12.1 was only tested on a subset of groups and visits because it was superseded by other variants of concern.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
fold rise | 10.84 [7.48 to 15.71] | 9.34 [5.48 to 15.92] | 11.84 [5.81 to 24.12] | 9.01 [5.38 to 15.10] | 8.65 [5.53 to 13.53]

16. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against BA.4/BA.5 in One Dose Groups.
Description: Pseudovirus Neutralization From Baseline Against BA.4/BA.5. Fold-rise is calculated by dividing post-vaccination results by the baseline value. The geometric mean of the fold rise is then reported.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
fold rise
  Day 15: number analyzed (Participants) | 27 | 25 | 26 | 25 | 26 | 0 | 0 | 0 | 1 | 0 | 0 | 46 | 49 | 50 | 100 | 100
  Day 15 | 12.31 [8.59 to 17.65] | 10.06 [6.42 to 15.77] | 16.19 [7.86 to 33.36] | 9.20 [5.26 to 16.09] | 12.25 [6.83 to 21.97] |  |  |  | 8.45 [NA to NA] — 95% confidence interval was not estimable as data from only 1 participant was analyzed |  |  | 3.10 [2.19 to 4.39] | 5.54 [3.64 to 8.44] | 4.37 [3.00 to 6.35] | 4.65 [3.76 to 5.77] | 8.04 [6.26 to 10.32]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 6.56 [5.11 to 8.42] | 10.34 [7.81 to 13.69] | 11.93 [8.98 to 15.84] | 8.45 [6.58 to 10.87] | 9.88 [7.45 to 13.11] | 4.21 [3.19 to 5.56] | 8.39 [5.88 to 11.98] | 9.51 [6.34 to 14.26] | 9.40 [6.76 to 13.07] | 9.72 [7.00 to 13.50] | 8.75 [5.73 to 13.37] | 3.68 [2.63 to 5.15] | 6.57 [4.15 to 10.41] | 5.46 [3.59 to 8.31] | 4.03 [3.25 to 5.00] | 6.64 [5.26 to 8.37]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 4.82 [3.48 to 6.67] | 8.98 [6.80 to 11.88] | 8.63 [6.31 to 11.81] | 6.64 [4.96 to 8.89] | 8.01 [5.80 to 11.08] | 3.96 [2.41 to 6.52] | 6.96 [4.54 to 10.67] | 6.65 [4.17 to 10.60] | 6.49 [4.22 to 9.97] | 6.55 [4.16 to 10.30] | 7.07 [4.28 to 11.67] | 3.22 [1.76 to 5.90] | 6.41 [3.73 to 11.02] | 4.81 [2.92 to 7.93] | 2.77 [2.17 to 3.54] | 5.27 [4.09 to 6.77]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 3.36 [2.31 to 4.88] | 6.08 [4.15 to 8.89] | 5.21 [3.58 to 7.58] | 5.29 [3.64 to 7.67] | 6.83 [4.57 to 10.21] | 5.80 [2.86 to 11.76] | 4.84 [2.88 to 8.15] | 4.92 [2.90 to 8.34] | 5.92 [3.65 to 9.62] | 5.07 [3.05 to 8.43] | 5.85 [3.25 to 10.53] | 5.39 [2.90 to 10.03] | 8.48 [4.54 to 15.84] | 6.86 [3.91 to 12.03] | 2.71 [2.04 to 3.60] | 4.34 [3.23 to 5.85]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 8.95 [6.10 to 13.13] | 11.67 [7.88 to 17.28] | 11.05 [7.58 to 16.12] | 9.92 [6.84 to 14.38] | 12.73 [8.47 to 19.13] | 10.41 [5.46 to 19.86] | 10.18 [6.23 to 16.62] | 7.00 [4.24 to 11.56] | 11.20 [6.32 to 19.82] | 9.77 [5.59 to 17.07] | 9.69 [5.40 to 17.37] | 8.60 [4.48 to 16.51] | 8.79 [4.94 to 15.66] | 8.53 [4.79 to 15.19] | 2.31 [1.67 to 3.18] | 3.24 [2.39 to 4.39]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 8.16 [5.60 to 11.90] | 10.49 [7.04 to 15.63] | 10.03 [6.87 to 14.64] | 8.47 [5.71 to 12.57] | 8.58 [5.75 to 12.79] | 10.05 [5.31 to 19.01] | 9.73 [5.70 to 16.61] | 6.70 [3.91 to 11.51] | 10.95 [6.04 to 19.86] | 13.41 [7.87 to 22.85] | 13.61 [7.24 to 25.58] | 7.36 [3.80 to 14.24] | 9.19 [5.23 to 16.16] | 8.73 [4.95 to 15.41] | 2.35 [1.68 to 3.28] | 2.88 [2.15 to 3.87]

17. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Pseudovirus Neutralization From Baseline Antibody Against BA.4/BA.5 in Two Dose Group.
Description: as for outcome 16
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
fold rise
  Day 15: number analyzed (Participants) | 1
  Day 15 | 40.80 [NA to NA] — 95% confidence interval is not estimable as data from only 1 participant was analyzed.
  Day 29: number analyzed (Participants) | 85
  Day 29 | 10.61 [8.04 to 14.00]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 8.51 [6.48 to 11.16]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 15.55 [11.70 to 20.67]
  Day 147 | 9.05 [6.56 to 12.48]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 11.11 [7.57 to 16.30]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 11.06 [7.23 to 16.92]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 11.68 [7.52 to 18.14]

18. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against Wa-1 in One Dose Groups.
Description: Geometric Mean (GM) AUC of Antibody Against Wa-1. The assay result, reported in arbitrary units, was repeated over a series of dilutions (e.g. 1/10, 1/100, 1/1000). These data were plotted, with dilution factor (1/dilution) on the x-axis and assay result on the y-axis, and the AUC was calculated as the area under the assay results from each dilution. As the x-axis of this AUC calculation was the dilution factor and the y-axis was the assay result in arbitrary units, the calculated AUC has units of arbitrary units*1/dilution.
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 98 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
Arbitrary Units*1/Dilution
  Day 1: number analyzed (Participants) | 98 | 111 | 100 | 99 | 96 | 49 | 52 | 53 | 51 | 50 | 52 | 47 | 48 | 52 | 100 | 100
  Day 1 | 160130.96 [129306.07 to 198304.11] | 207723.16 [175454.95 to 245925.88] | 202202.73 [166561.76 to 245470.18] | 196631.40 [163415.98 to 236598.09] | 212964.59 [175702.33 to 258129.29] | 235396.11 [173485.95 to 319399.50] | 182053.56 [142739.02 to 232196.48] | 170171.30 [126165.92 to 229525.31] | 165049.51 [123533.92 to 220517.08] | 187732.35 [147721.17 to 238580.79] | 225024.80 [172975.49 to 292736.06] | 232208.85 [174691.62 to 308663.64] | 207078.95 [151240.53 to 283533.07] | 223811.30 [162517.09 to 308222.95] | 216940.66 [179276.43 to 262517.77] | 227685.26 [191148.70 to 271205.49]
  Day 29: number analyzed (Participants) | 88 | 110 | 96 | 94 | 86 | 45 | 51 | 47 | 50 | 50 | 45 | 45 | 43 | 50 | 95 | 95
  Day 29 | 643473.03 [560692.10 to 738475.79] | 733522.42 [649743.77 to 828103.58] | 751245.45 [648796.71 to 869871.45] | 727260.22 [643219.99 to 822280.77] | 732226.74 [644366.79 to 832066.46] | 659275.24 [548924.63 to 791809.69] | 657238.13 [555813.86 to 777170.18] | 552682.55 [442382.31 to 690484.22] | 668859.02 [547609.32 to 816955.38] | 780465.85 [642036.37 to 948742.12] | 828997.70 [702454.95 to 978336.31] | 480315.31 [397529.55 to 580341.26] | 495494.62 [384679.35 to 638232.65] | 494440.20 [388582.83 to 629135.12] | 626852.32 [549349.76 to 715288.98] | 751965.51 [666099.41 to 848900.50]
  Day 91: number analyzed (Participants) | 91 | 108 | 94 | 93 | 91 | 47 | 49 | 48 | 47 | 46 | 48 | 45 | 45 | 50 | 97 | 96
  Day 91 | 438337.91 [378653.50 to 507429.94] | 491732.55 [427405.36 to 565741.40] | 514596.59 [432927.07 to 611672.65] | 500148.94 [442720.16 to 565027.27] | 536531.50 [457973.81 to 628564.44] | 548300.07 [447722.91 to 671471.03] | 461530.27 [376981.71 to 565041.19] | 391247.40 [303480.78 to 504396.12] | 448950.77 [358372.82 to 562422.10] | 514233.46 [410998.80 to 643398.59] | 556630.53 [454565.36 to 681612.76] | 398264.81 [307117.53 to 516463.06] | 428565.45 [340090.46 to 540057.33] | 438037.58 [339081.21 to 565873.06] | 442103.46 [380985.37 to 513026.18] | 510417.03 [444881.85 to 585606.14]
  Day 181: number analyzed (Participants) | 91 | 105 | 95 | 96 | 92 | 41 | 49 | 46 | 48 | 49 | 44 | 44 | 40 | 48 | 94 | 95
  Day 181 | 298887.11 [250797.08 to 356198.34] | 353554.44 [296724.80 to 421268.26] | 347652.35 [284713.04 to 424505.16] | 367923.35 [314484.84 to 430442.34] | 395234.07 [332468.37 to 469849.11] | 478836.67 [391278.37 to 585988.34] | 294887.23 [235836.33 to 368723.86] | 301817.71 [221380.26 to 411481.73] | 320772.07 [252468.56 to 407554.59] | 385153.46 [301669.57 to 491740.64] | 334355.35 [259649.52 to 430555.39] | 417943.47 [312516.72 to 558935.67] | 396620.26 [299395.40 to 525417.65] | 394207.59 [304879.45 to 509708.42] | 324842.08 [277309.16 to 380522.50] | 383432.41 [332019.90 to 442806.03]
  Day 271: number analyzed (Participants) | 90 | 96 | 90 | 95 | 87 | 40 | 49 | 48 | 46 | 47 | 48 | 44 | 42 | 45 | 87 | 94
  Day 271 | 390584.35 [325688.98 to 468410.50] | 431882.28 [367242.99 to 507898.89] | 452851.99 [382444.94 to 536220.79] | 475740.12 [400055.36 to 565743.35] | 466559.85 [387663.08 to 561513.61] | 580706.90 [476686.95 to 707425.50] | 346700.48 [276953.35 to 434012.52] | 301421.05 [218160.68 to 416457.49] | 394254.66 [298422.80 to 520860.80] | 421371.41 [321087.78 to 552976.09] | 383558.51 [285466.37 to 515357.13] | 442185.42 [342582.32 to 570747.33] | 414729.20 [300599.23 to 572191.43] | 394141.46 [291957.90 to 532088.67] | 271252.94 [226888.75 to 324291.80] | 286565.58 [245217.19 to 334886.11]
  Day 366: number analyzed (Participants) | 95 | 96 | 93 | 91 | 89 | 42 | 48 | 48 | 45 | 45 | 44 | 45 | 40 | 45 | 89 | 90
  Day 366 | 310610.18 [258096.07 to 373809.19] | 372637.70 [315316.19 to 440379.71] | 377586.71 [314604.53 to 453177.59] | 350750.36 [298128.48 to 412660.40] | 357990.63 [302163.02 to 424132.93] | 345763.94 [280205.28 to 426661.14] | 266067.35 [214976.08 to 329301.00] | 231315.61 [169652.11 to 315391.95] | 272137.87 [204275.55 to 362544.70] | 332233.81 [255504.78 to 432004.84] | 303821.76 [226449.66 to 407629.93] | 319747.17 [243868.05 to 419235.93] | 281475.15 [206656.68 to 383381.07] | 301625.72 [225119.59 to 404132.20] | 239959.56 [201762.03 to 285388.63] | 242634.48 [207407.30 to 283844.85]

19. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against Wa-1 in Two Dose Group.
Description: as for outcome 18
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
Arbitrary Units*1/Dilution
  Day 1: number analyzed (Participants) | 85
  Day 1 | 170503.26 [137457.73 to 211493.11]
  Day 29: number analyzed (Participants) | 77
  Day 29 | 606554.56 [517874.98 to 710419.40]
  Day 57: number analyzed (Participants) | 79
  Day 57 | 494683.51 [420526.83 to 581917.14]
  Day 85: number analyzed (Participants) | 77
  Day 85 | 762319.06 [664514.22 to 874519.05]
  Day 147: number analyzed (Participants) | 78
  Day 147 | 582298.62 [491139.17 to 690378.01]
  Day 237: number analyzed (Participants) | 82
  Day 237 | 447713.57 [368540.63 to 543895.11]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 395463.67 [327719.15 to 477212.02]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 302772.82 [249170.24 to 367906.61]

20. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against B.1.351 in One Dose Groups.
Description: Geometric Mean (GM) AUC of Antibody Against B.1.351. The assay result, reported in arbitrary units, was repeated over a series of dilutions (e.g. 1/10, 1/100, 1/1000). These data were plotted, with dilution factor (1/dilution) on the x-axis and assay result on the y-axis, and the AUC was calculated as the area under the assay results from each dilution. As the x-axis of this AUC calculation was the dilution factor and the y-axis was the assay result in arbitrary units, the calculated AUC has units of arbitrary units*1/dilution.
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
Arbitrary Units*1/Dilution
  Day 1: number analyzed (Participants) | 99 | 113 | 100 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 52 | 48 | 49 | 52 | 100 | 100
  Day 1 | 93551.19 [75078.90 to 116568.38] | 129906.22 [109275.29 to 154432.23] | 116649.05 [95341.67 to 142718.31] | 115206.13 [95211.58 to 139399.56] | 128531.47 [104670.04 to 157832.56] | 135763.15 [99440.49 to 185353.40] | 104424.42 [80261.61 to 135861.47] | 110265.46 [80618.46 to 150814.99] | 100277.89 [74167.67 to 135580.02] | 121192.68 [91029.66 to 161350.31] | 135028.37 [102158.31 to 178474.58] | 150238.68 [108957.54 to 207160.17] | 134064.73 [95854.88 to 187505.86] | 139963.38 [100342.92 to 195227.99] | 136025.14 [111826.03 to 165460.93] | 144727.88 [120097.52 to 174409.60]
  Day 29: number analyzed (Participants) | 96 | 110 | 94 | 93 | 91 | 48 | 49 | 49 | 50 | 47 | 46 | 46 | 44 | 50 | 98 | 95
  Day 29 | 436540.44 [376880.27 to 505644.81] | 536040.87 [474391.87 to 605701.39] | 497454.13 [424663.31 to 582721.91] | 522838.44 [461094.90 to 592849.84] | 510066.75 [439438.66 to 592046.44] | 468813.37 [381774.62 to 575695.62] | 499652.43 [416521.98 to 599374.26] | 441732.81 [352523.10 to 553517.97] | 536875.49 [434894.96 to 662769.91] | 535912.15 [434670.77 to 660734.18] | 590251.89 [493880.47 to 705428.37] | 327932.05 [263367.44 to 408324.69] | 386837.28 [294054.43 to 508895.86] | 359000.12 [276299.54 to 466454.22] | 479928.00 [418836.28 to 549930.61] | 547431.70 [482946.41 to 620527.36]
  Day 91: number analyzed (Participants) | 91 | 110 | 96 | 97 | 94 | 48 | 50 | 49 | 48 | 49 | 49 | 47 | 47 | 51 | 98 | 97
  Day 91 | 260600.97 [224396.48 to 302646.74] | 353154.19 [307127.09 to 406079.06] | 337018.67 [279601.80 to 406226.21] | 368777.24 [323248.64 to 420718.39] | 364466.11 [307829.74 to 431522.78] | 343409.80 [275950.45 to 427360.39] | 339016.33 [274108.66 to 419293.84] | 304500.86 [233667.50 to 396806.47] | 358322.49 [282483.03 to 454522.90] | 395543.34 [310803.13 to 503387.91] | 396620.95 [318981.99 to 493156.94] | 264515.83 [200295.28 to 349327.37] | 315462.53 [244506.65 to 407009.83] | 296474.19 [226058.64 to 388823.64] | 307530.83 [262787.72 to 359892.04] | 360330.74 [312470.31 to 415521.85]
  Day 181: number analyzed (Participants) | 91 | 105 | 97 | 96 | 94 | 41 | 49 | 47 | 50 | 50 | 45 | 44 | 41 | 49 | 94 | 94
  Day 181 | 173909.68 [143380.99 to 210938.54] | 237513.05 [199090.53 to 283350.74] | 228919.38 [183497.82 to 285584.22] | 238062.10 [203710.45 to 278206.46] | 258839.20 [214625.36 to 312161.32] | 303657.19 [245914.64 to 374958.11] | 192668.11 [150365.03 to 246872.57] | 219015.58 [159282.21 to 301149.93] | 245072.17 [187309.29 to 320648.11] | 263281.28 [201601.41 to 343832.08] | 234800.63 [178900.06 to 308168.36] | 275654.28 [204726.77 to 371154.58] | 300882.56 [221725.62 to 408298.85] | 287091.71 [217849.16 to 378342.73] | 235298.55 [198020.37 to 279594.51] | 280572.85 [240451.74 to 327388.45]
  Day 271: number analyzed (Participants) | 89 | 98 | 90 | 96 | 88 | 41 | 49 | 49 | 46 | 47 | 49 | 44 | 41 | 45 | 87 | 94
  Day 271 | 258643.48 [212437.89 to 314898.85] | 328407.16 [276854.00 to 389560.08] | 331083.82 [275761.38 to 397504.89] | 336408.76 [281631.43 to 401840.29] | 338933.50 [278671.06 to 412227.66] | 408169.15 [330873.40 to 503522.05] | 242648.32 [188718.40 to 311989.76] | 222230.23 [160616.45 to 307479.57] | 294022.31 [219359.96 to 394097.09] | 311998.19 [231177.80 to 421073.61] | 284552.50 [209437.76 to 386607.11] | 315964.73 [242926.24 to 410963.04] | 312951.39 [222960.86 to 439263.50] | 300475.72 [217340.28 to 415411.53] | 190613.29 [157623.37 to 230507.85] | 199914.23 [169853.36 to 235295.30]
  Day 366: number analyzed (Participants) | 89 | 101 | 94 | 95 | 90 | 44 | 48 | 48 | 46 | 47 | 46 | 46 | 40 | 45 | 89 | 90
  Day 366 | 221467.29 [180356.70 to 271948.65] | 288113.03 [239895.57 to 346021.90] | 267894.35 [219924.61 to 326327.20] | 249713.10 [209280.07 to 297957.82] | 247236.94 [206166.46 to 296489.08] | 243160.36 [192000.49 to 307952.15] | 181309.72 [143792.20 to 228616.12] | 156958.86 [116124.63 to 212152.10] | 200084.98 [148201.09 to 270132.95] | 253664.70 [187302.66 to 343539.07] | 231244.70 [170470.44 to 313685.55] | 227063.40 [167501.42 to 307805.08] | 216318.74 [154124.59 to 303610.19] | 215517.27 [158858.38 to 292384.30] | 164587.63 [136637.76 to 198254.78] | 163821.61 [139478.93 to 192412.70]

21. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against B.1.351 in Two Dose Group.
Description: as for outcome 20
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
Arbitrary Units*1/Dilution
  Day 1: number analyzed (Participants) | 85
  Day 1 | 99752.03 [79297.68 to 125482.45]
  Day 29: number analyzed (Participants) | 78
  Day 29 | 467456.52 [396238.18 to 551475.38]
  Day 57: number analyzed (Participants) | 80
  Day 57 | 383162.27 [321719.82 to 456339.08]
  Day 85: number analyzed (Participants) | 77
  Day 85 | 601632.71 [518559.18 to 698014.67]
  Day 147: number analyzed (Participants) | 83
  Day 147 | 440762.25 [368674.52 to 526945.44]
  Day 237 | 339450.17 [277014.51 to 415958.07]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 290896.60 [238344.40 to 355035.95]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 217113.45 [176796.73 to 266623.98]

22. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against BA.1 in One Dose Groups.
Description: Geometric Mean (GM) AUC of Antibody Against BA.1. The assay result, reported in arbitrary units, was repeated over a series of dilutions (e.g. 1/10, 1/100, 1/1000). These data were plotted, with dilution factor (1/dilution) on the x-axis and assay result on the y-axis, and the AUC was calculated as the area under the assay results from each dilution. As the x-axis of this AUC calculation was the dilution factor and the y-axis was the assay result in arbitrary units, the calculated AUC has units of arbitrary units*1/dilution.
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
Arbitrary Units*1/Dilution
  Day 1 | 35858.62 [28544.50 to 45046.88] | 50667.27 [41821.05 to 61384.70] | 46101.27 [36611.11 to 58051.43] | 43880.60 [35811.70 to 53767.55] | 48636.02 [39357.99 to 60101.20] | 53148.74 [38023.65 to 74290.30] | 37332.20 [28270.98 to 49297.67] | 39668.84 [28557.73 to 55103.00] | 36466.06 [26603.75 to 49984.44] | 46523.96 [34272.24 to 63155.46] | 56154.79 [40714.86 to 77449.85] | 55708.69 [39647.52 to 78276.23] | 51579.87 [35935.37 to 74035.22] | 53338.07 [37253.33 to 76367.68] | 48508.52 [39245.75 to 59957.49] | 50242.30 [41180.19 to 61298.62]
  Day 29: number analyzed (Participants) | 97 | 112 | 99 | 98 | 93 | 48 | 51 | 50 | 50 | 51 | 52 | 46 | 46 | 51 | 99 | 98
  Day 29 | 191702.35 [164106.87 to 223938.16] | 245795.04 [214464.11 to 281703.09] | 243857.48 [202010.59 to 294373.04] | 268727.94 [229848.03 to 314184.58] | 245471.75 [209505.23 to 287612.76] | 199576.30 [159461.92 to 249781.88] | 228987.60 [183030.45 to 286484.14] | 216259.20 [166594.92 to 280729.10] | 215235.97 [171659.19 to 269874.99] | 253784.67 [197499.84 to 326109.93] | 343044.44 [271270.81 to 433808.14] | 140177.75 [111549.63 to 176153.01] | 168689.34 [122859.78 to 231614.39] | 152376.48 [113422.48 to 204708.92] | 219690.36 [188573.15 to 255942.36] | 242501.72 [208975.92 to 281406.04]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 111776.32 [94301.82 to 132488.92] | 150303.44 [128509.07 to 175794.00] | 154578.88 [124948.41 to 191235.97] | 168167.22 [144346.78 to 195918.55] | 163330.96 [134898.13 to 197756.65] | 130887.24 [104132.56 to 164515.98] | 131524.99 [104482.91 to 165566.05] | 138870.07 [102534.27 to 188082.45] | 142416.99 [108517.33 to 186906.53] | 165935.22 [126207.83 to 218167.89] | 174816.63 [138986.83 to 219883.08] | 108504.45 [80492.50 to 146264.74] | 119334.36 [90217.56 to 157848.32] | 110503.80 [83053.87 to 147026.12] | 131000.91 [110029.50 to 155969.42] | 140386.22 [119592.54 to 164795.31]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 45 | 43 | 50 | 94 | 95
  Day 181 | 67934.34 [55305.96 to 83446.24] | 95644.75 [79114.54 to 115628.79] | 89619.90 [70683.74 to 113629.07] | 96998.27 [81579.63 to 115331.05] | 103752.38 [85159.85 to 126404.14] | 117299.54 [92895.44 to 148114.72] | 78601.03 [59970.15 to 103019.95] | 96217.34 [68381.48 to 135384.29] | 88377.85 [67626.56 to 115496.69] | 100149.77 [76233.87 to 131568.49] | 108679.49 [78803.64 to 149881.79] | 106506.21 [77882.34 to 145650.13] | 122787.89 [84823.97 to 177742.99] | 107521.40 [78962.21 to 146409.93] | 93570.97 [77636.77 to 112775.52] | 102367.44 [86226.19 to 121530.27]
  Day 271: number analyzed (Participants) | 90 | 100 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 45 | 43 | 47 | 87 | 94
  Day 271 | 99192.03 [80277.18 to 122563.58] | 131888.79 [109150.10 to 159364.50] | 139325.91 [113298.48 to 171332.48] | 139410.13 [114786.42 to 169316.06] | 139473.50 [112336.10 to 173166.57] | 149877.01 [120234.22 to 186827.99] | 95340.03 [72516.76 to 125346.49] | 92710.85 [66119.63 to 129996.20] | 112221.17 [81586.64 to 154358.50] | 122393.65 [89820.97 to 166778.48] | 122432.06 [87816.74 to 170691.93] | 127066.31 [95295.52 to 169429.24] | 120389.82 [82167.30 to 176392.65] | 117354.27 [81343.60 to 169306.81] | 70720.41 [56789.58 to 88068.56] | 66434.87 [55341.74 to 79751.60]
  Day 366: number analyzed (Participants) | 89 | 100 | 95 | 95 | 90 | 44 | 48 | 49 | 48 | 47 | 47 | 46 | 39 | 45 | 89 | 90
  Day 366 | 79561.28 [63948.44 to 98985.96] | 105460.05 [86839.37 to 128073.50] | 106503.48 [85253.96 to 133049.43] | 99354.35 [81713.17 to 120804.13] | 92964.28 [76395.58 to 113126.41] | 85243.80 [66428.02 to 109389.15] | 67777.11 [52510.16 to 87482.81] | 63755.85 [45948.96 to 88463.56] | 78292.70 [55674.78 to 110099.19] | 95692.23 [69900.64 to 131000.28] | 97653.95 [69113.30 to 137980.58] | 78559.42 [57473.61 to 107381.14] | 70561.84 [48140.57 to 103425.72] | 76460.37 [54315.81 to 107633.26] | 61045.92 [49522.11 to 75251.32] | 54849.37 [45941.98 to 65483.76]

23. Primary Outcome: Geometric Mean (GM) AUC of Antibody Against BA.1 in Two Dose Group.
Description: as for outcome 22
Time Frame: Day 1 Pre-Booster Dose, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units*1/Dilution
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
Arbitrary Units*1/Dilution
  Day 1 | 39029.80 [30219.86 to 50408.08]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 232195.94 [191647.37 to 281323.74]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 184155.65 [150366.02 to 225538.33]
  Day 85: number analyzed (Participants) | 83
  Day 85 | 303406.48 [255832.11 to 359827.76]
  Day 147 | 206168.23 [167818.87 to 253281.06]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 132219.79 [106176.30 to 164651.37]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 112933.35 [91545.00 to 139318.83]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 79707.84 [63831.66 to 99532.74]

24. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
titer
  Day 1 | 3245.3 [2437.1 to 4321.7] | 3959.5 [3011.8 to 5205.5] | 3537.5 [2621.4 to 4773.8] | 3874.1 [2930.3 to 5121.8] | 3595.9 [2603.1 to 4967.3] | 4761.5 [3136.8 to 7227.9] | 3720.3 [2462.4 to 5620.8] | 3982.2 [2757.9 to 5750.0] | 3687.5 [2246.9 to 6051.6] | 4423.3 [3121.8 to 6267.3] | 4686.6 [3120.4 to 7039.0] | 5196.7 [3499.0 to 7718.1] | 3432.5 [1970.0 to 5980.5] | 5419.9 [3586.6 to 8190.4] | 7448.8 [5944.6 to 9333.5] | 7786.8 [6056.9 to 10010.7]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 21060.3 [17431.9 to 25443.9] | 21523.4 [17685.7 to 26194.0] | 24323.2 [19090.6 to 30989.9] | 19304.9 [16023.6 to 23258.2] | 26279.7 [21858.1 to 31595.7] | 21566.8 [16564.3 to 28080.0] | 14986.8 [10502.8 to 21385.1] | 15842.2 [11653.3 to 21536.8] | 18854.6 [13408.9 to 26512.1] | 22458.9 [17223.2 to 29286.4] | 28322.2 [21912.1 to 36607.4] | 8102.7 [5946.9 to 11040.1] | 9670.5 [7151.0 to 13077.7] | 9982.9 [7470.3 to 13340.7] | 27493.0 [23775.4 to 31791.9] | 33715.5 [29188.9 to 38944.1]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 15972.1 [13059.2 to 19534.7] | 16815.7 [13977.3 to 20230.6] | 18250.6 [14438.1 to 23069.8] | 14380.9 [11875.8 to 17414.4] | 17680.2 [13979.4 to 22360.7] | 16440.9 [12881.8 to 20983.4] | 15825.6 [12730.1 to 19673.9] | 15451.6 [11369.0 to 21000.3] | 15674.6 [11193.5 to 21949.7] | 19718.1 [14861.3 to 26162.3] | 24139.0 [18398.1 to 31671.2] | 10390.1 [7637.2 to 14135.4] | 13898.2 [9838.0 to 19634.0] | 14825.3 [10909.1 to 20147.4] | 31502.1 [26665.9 to 37215.4] | 36372.7 [30960.4 to 42731.2]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 11701.1 [8786.7 to 15582.2] | 14410.2 [11561.7 to 17960.4] | 16558.4 [12500.4 to 21933.6] | 14296.6 [11443.9 to 17860.4] | 16567.5 [13410.8 to 20467.1] | 8878.3 [6899.7 to 11424.3] | 7168.4 [4916.7 to 10451.4] | 8157.4 [5738.9 to 11595.1] | 8344.8 [5632.6 to 12363.1] | 10091.6 [7429.1 to 13708.3] | 11463.3 [8532.4 to 15400.8] | 11464.2 [8344.3 to 15750.7] | 12503.4 [9048.2 to 17278.0] | 11949.2 [8770.5 to 16280.0] | 14685.9 [12121.8 to 17792.3] | 18941.5 [15945.2 to 22500.8]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 6903.6 [5136.3 to 9279.0] | 7562.1 [5654.8 to 10112.8] | 8909.5 [6694.5 to 11857.3] | 7621.8 [5919.8 to 9813.1] | 9964.2 [7705.7 to 12884.7] | 13012.4 [9511.7 to 17801.4] | 6369.6 [4220.6 to 9613.0] | 7294.8 [5036.4 to 10565.9] | 7954.9 [5434.1 to 11644.9] | 9107.1 [6525.4 to 12710.2] | 10985.5 [7501.6 to 16087.3] | 12634.3 [8474.3 to 18836.5] | 10278.3 [6394.0 to 16522.4] | 13441.8 [9717.9 to 18592.7] | 11401.6 [9285.0 to 14000.7] | 12407.1 [9795.0 to 15715.9]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 11298.3 [8553.7 to 14923.5] | 12807.0 [10031.3 to 16350.8] | 12567.4 [9669.8 to 16333.4] | 11943.9 [9633.0 to 14809.2] | 12712.9 [9740.9 to 16591.7] | 15654.4 [11271.3 to 21741.9] | 7715.8 [5167.5 to 11520.9] | 7211.2 [4925.9 to 10556.8] | 10557.7 [7065.3 to 15776.5] | 9559.5 [6174.7 to 14799.9] | 10701.5 [6765.3 to 16928.0] | 12557.1 [8887.5 to 17741.8] | 10729.0 [7461.8 to 15426.7] | 13065.9 [9274.8 to 18406.7] | 9755.4 [7882.1 to 12073.9] | 10562.7 [8377.0 to 13318.6]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 8671.6 [6723.5 to 11184.1] | 8756.9 [6440.1 to 11907.3] | 8552.4 [6376.5 to 11470.6] | 8065.4 [6207.8 to 10478.8] | 9784.4 [7382.6 to 12967.6] | 13214.9 [9643.9 to 18108.1] | 7644.9 [5080.0 to 11504.8] | 6661.2 [4285.1 to 10354.8] | 9652.1 [6186.6 to 15059.1] | 12279.8 [8351.9 to 18054.8] | 12341.7 [8245.4 to 18473.2] | 13314.0 [9596.9 to 18470.8] | 10449.0 [7002.5 to 15591.9] | 14255.0 [9505.4 to 21377.9] | 8366.7 [6770.6 to 10339.1] | 8509.6 [6732.7 to 10755.6]

25. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G in Two Dose Group.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
titer
  Day 1 | 3358.3 [2495.4 to 4519.7]
  Day 15 | 17962.2 [13481.6 to 23932.0]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 12816.7 [9298.0 to 17667.2]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 11171.5 [8416.8 to 14827.9]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 16328.8 [12496.7 to 21335.9]
  Day 147 | 9988.4 [7645.1 to 13050.0]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 12128.0 [9225.4 to 15943.8]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 8859.3 [6651.5 to 11799.9]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 10156.6 [7417.9 to 13906.4]

26. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351 in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
titer
  Day 1 | 810.8 [575.1 to 1143.2] | 1069.4 [791.3 to 1445.1] | 862.6 [609.1 to 1221.6] | 933.8 [648.2 to 1345.2] | 963.6 [682.3 to 1360.8] | 1223.6 [705.0 to 2123.6] | 1056.9 [630.2 to 1772.2] | 922.8 [549.7 to 1548.9] | 977.0 [583.6 to 1635.6] | 1183.1 [730.7 to 1915.5] | 1065.4 [617.0 to 1839.6] | 1426.0 [805.6 to 2524.0] | 863.5 [453.6 to 1643.8] | 1556.0 [885.9 to 2732.7] | 2821.0 [2160.5 to 3683.3] | 2871.5 [2143.5 to 3846.8]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 7678.4 [6047.9 to 9748.5] | 13422.2 [10731.1 to 16788.1] | 9926.8 [7393.7 to 13327.9] | 11214.3 [8583.3 to 14651.8] | 10820.3 [8304.5 to 14098.3] | 7611.7 [5395.7 to 10737.7] | 8476.8 [5772.1 to 12449.0] | 8830.1 [6233.6 to 12508.2] | 10447.5 [7092.5 to 15389.3] | 9901.1 [7124.1 to 13760.6] | 11367.9 [7962.3 to 16230.0] | 2849.5 [1917.7 to 4233.9] | 5099.4 [3623.4 to 7176.6] | 5075.6 [3582.4 to 7191.2] | 15520.2 [12922.7 to 18639.9] | 19051.8 [15893.6 to 22837.4]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 4815.7 [3673.9 to 6312.4] | 9771.6 [7840.6 to 12178.0] | 6919.2 [5121.9 to 9347.2] | 7551.7 [5771.2 to 9881.6] | 6790.7 [5021.5 to 9183.2] | 5266.4 [3842.1 to 7218.6] | 7961.0 [5445.0 to 11639.5] | 8652.2 [6017.6 to 12440.2] | 9007.8 [6131.2 to 13234.0] | 8014.2 [5812.4 to 11050.1] | 9167.2 [6353.9 to 13226.3] | 4081.5 [2773.6 to 6006.1] | 8285.2 [5408.7 to 12691.3] | 8103.0 [5628.4 to 11665.6] | 13674.7 [10962.7 to 17057.6] | 16252.8 [13337.6 to 19805.1]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 3575.3 [2573.1 to 4967.7] | 7029.6 [5367.1 to 9207.0] | 5685.7 [4010.9 to 8059.8] | 6703.6 [4998.4 to 8990.5] | 6534.1 [4915.0 to 8686.5] | 2742.8 [1842.9 to 4081.9] | 3778.1 [2490.6 to 5731.3] | 4135.7 [2700.0 to 6334.9] | 4507.0 [2907.1 to 6987.4] | 4316.6 [3000.1 to 6210.6] | 4879.2 [3250.9 to 7323.0] | 4194.0 [2779.8 to 6327.6] | 6814.3 [4711.6 to 9855.5] | 5876.1 [3975.4 to 8685.5] | 6168.0 [4943.1 to 7696.4] | 7758.5 [6231.9 to 9658.9]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 2033.2 [1443.9 to 2863.0] | 3466.0 [2460.9 to 4881.5] | 2804.2 [1905.6 to 4126.7] | 3370.8 [2516.2 to 4515.6] | 4008.9 [3015.1 to 5330.2] | 4110.3 [2739.6 to 6166.9] | 2625.3 [1710.6 to 4029.0] | 2624.9 [1628.1 to 4231.9] | 3150.5 [2069.5 to 4796.0] | 2791.2 [1821.5 to 4277.2] | 3566.1 [2122.6 to 5991.3] | 4227.2 [2765.5 to 6461.3] | 4814.4 [2895.5 to 8004.8] | 6141.5 [4216.7 to 8944.9] | 5741.9 [4433.6 to 7436.3] | 6041.1 [4629.0 to 7884.1]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 3423.4 [2387.2 to 4909.3] | 5039.4 [3659.0 to 6940.6] | 3938.1 [2854.8 to 5432.4] | 4442.3 [3348.2 to 5893.9] | 4766.7 [3544.9 to 6409.7] | 7104.4 [4649.9 to 10854.5] | 4105.5 [2634.2 to 6398.6] | 3133.2 [1992.4 to 4927.1] | 4943.1 [3054.2 to 8000.3] | 4537.9 [2802.9 to 7346.8] | 5236.9 [3117.4 to 8797.4] | 5853.2 [4080.6 to 8395.6] | 6449.5 [4256.0 to 9773.5] | 7143.7 [4754.8 to 10732.7] | 3588.4 [2776.1 to 4638.3] | 3622.5 [2819.5 to 4654.4]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 2857.4 [2084.8 to 3916.4] | 3796.1 [2709.6 to 5318.1] | 2829.1 [2003.5 to 3994.9] | 3126.2 [2305.1 to 4239.7] | 3498.5 [2497.4 to 4900.8] | 4782.9 [3210.1 to 7126.3] | 3221.4 [2083.5 to 4980.7] | 2377.1 [1522.8 to 3710.6] | 4056.6 [2538.9 to 6481.6] | 3906.0 [2435.9 to 6263.4] | 4325.9 [2713.3 to 6897.2] | 4472.8 [3134.2 to 6383.2] | 3796.0 [2222.7 to 6483.0] | 5337.7 [3410.3 to 8354.5] | 4041.5 [3153.9 to 5178.8] | 4026.9 [3119.8 to 5197.9]

27. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351 in Two Dose Group.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
titer
  Day 1 | 847.0 [583.8 to 1228.9]
  Day 15 | 11275.7 [8306.0 to 15307.1]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 7800.2 [5548.0 to 10966.6]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 6008.9 [4426.1 to 8157.6]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 10285.2 [7694.0 to 13749.1]
  Day 147 | 5061.1 [3755.3 to 6821.1]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 5362.8 [3812.3 to 7543.9]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 4295.6 [3036.0 to 6078.0]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 3780.4 [2636.4 to 5420.9]

28. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.617.2 in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.617.2.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
titer
  Day 1 | 1602.4 [1174.8 to 2185.7] | 1842.0 [1373.9 to 2469.6] | 1783.4 [1316.2 to 2416.4] | 1898.6 [1430.1 to 2520.6] | 1771.4 [1279.3 to 2453.0] | 2261.3 [1434.3 to 3565.0] | 1753.6 [1107.8 to 2775.8] | 1775.8 [1171.4 to 2692.2] | 1849.3 [1125.3 to 3039.1] | 2232.5 [1526.5 to 3265.1] | 2032.3 [1330.4 to 3104.6] | 2679.5 [1774.8 to 4045.4] | 1750.1 [1001.0 to 3059.8] | 2493.9 [1537.8 to 4044.4] | 3315.7 [2635.0 to 4172.1] | 3637.2 [2844.8 to 4650.3]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 11566.9 [9470.4 to 14127.6] | 13447.7 [10965.6 to 16491.6] | 14581.1 [11343.1 to 18743.3] | 11575.4 [9504.5 to 14097.4] | 13975.9 [11085.6 to 17619.8] | 10868.1 [8185.9 to 14429.0] | 8689.0 [6094.6 to 12387.8] | 8705.4 [6258.6 to 12109.0] | 9519.2 [6726.2 to 13472.1] | 12004.8 [9161.0 to 15731.3] | 13331.1 [9916.6 to 17921.3] | 3666.9 [2627.6 to 5117.3] | 5005.2 [3636.1 to 6889.9] | 4820.9 [3611.4 to 6435.5] | 14610.6 [12510.1 to 17063.9] | 18199.3 [15594.2 to 21239.6]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 7899.3 [6367.4 to 9799.7] | 9742.0 [7994.1 to 11872.1] | 11005.1 [8637.1 to 14022.2] | 8256.2 [6796.3 to 10029.6] | 9696.2 [7590.3 to 12386.3] | 8444.4 [6585.2 to 10828.4] | 9095.1 [7075.8 to 11690.5] | 8504.4 [6009.9 to 12034.2] | 9067.6 [6354.4 to 12939.3] | 10754.4 [7991.5 to 14472.5] | 11738.3 [8902.5 to 15477.4] | 5768.5 [4208.2 to 7907.3] | 8746.4 [6041.2 to 12663.0] | 8863.7 [6491.9 to 12102.0] | 13482.3 [11287.1 to 16104.5] | 16409.4 [13763.9 to 19563.5]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 5329.5 [3999.3 to 7102.1] | 7977.7 [6321.4 to 10068.0] | 8256.9 [6229.2 to 10944.7] | 7267.3 [5609.0 to 9415.7] | 8651.8 [6889.2 to 10865.3] | 4874.8 [3636.6 to 6534.5] | 4253.7 [2920.9 to 6194.6] | 4854.3 [3328.6 to 7079.3] | 4709.7 [3141.7 to 7060.2] | 5475.8 [4076.3 to 7355.8] | 6208.7 [4502.6 to 8561.1] | 5543.9 [3922.4 to 7835.6] | 7065.7 [5057.1 to 9872.3] | 6475.1 [4668.5 to 8981.0] | 6349.1 [5282.5 to 7631.0] | 8184.0 [6789.8 to 9864.5]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 2933.9 [2183.6 to 3942.0] | 3564.8 [2637.9 to 4817.4] | 3824.7 [2824.2 to 5179.6] | 3499.3 [2740.4 to 4468.5] | 4143.8 [3140.3 to 5468.1] | 5684.5 [4062.5 to 7954.1] | 2797.9 [1901.6 to 4116.6] | 3337.3 [2232.2 to 4989.5] | 3323.3 [2224.6 to 4964.6] | 4026.4 [2909.5 to 5572.0] | 4109.5 [2657.3 to 6355.5] | 4968.0 [3436.3 to 7182.4] | 5343.6 [3331.9 to 8569.9] | 6290.0 [4603.3 to 8594.8] | 5798.8 [4722.9 to 7119.7] | 6884.7 [5448.9 to 8698.9]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 4773.6 [3608.9 to 6314.1] | 5270.2 [3985.1 to 6969.7] | 4992.4 [3750.8 to 6645.1] | 5022.5 [3971.7 to 6351.3] | 5294.9 [4064.0 to 6898.7] | 7566.2 [5348.9 to 10702.8] | 3649.7 [2459.8 to 5415.4] | 3360.2 [2234.3 to 5053.6] | 4730.2 [3074.0 to 7278.8] | 4792.7 [3112.0 to 7381.2] | 5104.3 [3208.7 to 8119.7] | 6223.0 [4405.2 to 8791.0] | 5963.9 [4020.2 to 8847.4] | 6591.1 [4608.9 to 9425.8] | 4604.6 [3741.6 to 5666.7] | 5006.9 [3957.9 to 6334.0]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 3949.6 [3028.8 to 5150.3] | 4289.1 [3093.2 to 5947.3] | 4011.9 [2968.1 to 5422.8] | 3690.3 [2835.2 to 4803.3] | 4186.9 [3078.7 to 5694.0] | 6333.9 [4596.5 to 8727.9] | 3663.3 [2440.5 to 5498.7] | 3161.0 [2058.7 to 4853.5] | 4490.3 [2921.9 to 6900.5] | 5671.3 [3836.8 to 8382.7] | 5700.1 [3730.7 to 8709.1] | 5301.9 [3793.0 to 7410.9] | 4295.2 [2611.0 to 7065.8] | 6388.3 [4296.9 to 9497.8] | 5333.6 [4300.9 to 6614.3] | 5745.6 [4521.9 to 7300.6]

29. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.617.2 in Two Dose Group.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.617.2.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
titer
  Day 1 | 1508.5 [1079.6 to 2107.8]
  Day 15 | 10135.8 [7387.8 to 13905.9]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 7478.5 [5461.1 to 10241.1]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 6256.1 [4713.1 to 8304.1]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 9866.0 [7520.7 to 12942.7]
  Day 147 | 5012.4 [3723.0 to 6748.3]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 5004.8 [3673.2 to 6819.2]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 3856.0 [2814.3 to 5283.2]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 3919.6 [2825.7 to 5437.0]

30. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.1 in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.1.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
titer
  Day 1 | 264.4 [185.4 to 377.1] | 311.2 [222.9 to 434.5] | 278.1 [194.3 to 397.9] | 343.8 [237.8 to 497.0] | 348.4 [241.3 to 503.1] | 420.3 [230.7 to 765.9] | 306.8 [177.1 to 531.6] | 329.8 [197.2 to 551.4] | 271.2 [156.9 to 468.8] | 360.2 [207.2 to 626.2] | 346.4 [189.2 to 634.0] | 413.6 [227.3 to 752.7] | 291.6 [154.4 to 550.7] | 366.2 [207.0 to 647.8] | 1103.1 [838.7 to 1450.9] | 1002.9 [727.4 to 1382.7]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 2669.9 [2028.0 to 3515.0] | 5278.9 [4017.1 to 6936.9] | 4544.2 [3339.9 to 6182.6] | 6014.6 [4656.4 to 7768.9] | 5339.3 [4039.5 to 7057.3] | 2662.2 [1806.4 to 3923.5] | 3753.3 [2543.2 to 5539.3] | 4781.7 [3304.3 to 6919.5] | 3315.5 [2140.0 to 5136.6] | 3570.4 [2507.8 to 5083.3] | 5544.3 [3788.8 to 8113.1] | 1221.8 [796.0 to 1875.6] | 1966.6 [1309.5 to 2953.5] | 1636.0 [1067.1 to 2508.2] | 6558.3 [5249.4 to 8193.5] | 6511.2 [5112.8 to 8291.9]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 97 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 1863.8 [1438.3 to 2415.2] | 3967.2 [3043.9 to 5170.7] | 3320.9 [2447.7 to 4505.8] | 3994.1 [3081.7 to 5176.6] | 3520.8 [2585.9 to 4793.7] | 1602.1 [1100.9 to 2331.6] | 2532.9 [1705.8 to 3761.0] | 3852.6 [2721.7 to 5453.2] | 2301.1 [1549.8 to 3416.7] | 2547.3 [1788.9 to 3627.2] | 3285.6 [2210.9 to 4882.7] | 1071.7 [644.2 to 1783.0] | 2367.4 [1475.1 to 3799.4] | 1824.4 [1151.5 to 2890.6] | 5211.8 [4210.1 to 6451.9] | 5056.7 [3935.1 to 6498.1]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 1095.3 [804.3 to 1491.7] | 2492.5 [1850.4 to 3357.5] | 2234.9 [1604.1 to 3113.7] | 2382.6 [1754.9 to 3234.8] | 2460.1 [1766.4 to 3426.1] | 1228.7 [796.7 to 1894.8] | 1851.5 [1151.8 to 2976.2] | 3011.7 [2016.3 to 4498.4] | 1728.7 [1064.2 to 2808.3] | 1895.6 [1228.8 to 2924.1] | 2726.7 [1732.5 to 4291.4] | 1247.1 [798.4 to 1947.9] | 1756.6 [1117.6 to 2760.8] | 1471.8 [874.5 to 2477.2] | 3954.1 [3130.7 to 4994.0] | 3963.2 [3131.0 to 5016.5]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 741.1 [512.2 to 1072.5] | 1583.8 [1125.1 to 2229.5] | 1226.9 [833.8 to 1805.4] | 1634.9 [1197.4 to 2232.2] | 1721.4 [1248.5 to 2373.3] | 1801.7 [1137.3 to 2854.0] | 1214.8 [728.5 to 2025.7] | 1859.4 [1174.6 to 2943.6] | 1299.1 [815.5 to 2069.6] | 1413.4 [876.4 to 2279.3] | 2021.5 [1183.2 to 3453.7] | 1939.9 [1249.8 to 3011.1] | 2541.8 [1484.8 to 4351.3] | 2310.1 [1527.5 to 3493.8] | 3361.6 [2601.1 to 4344.6] | 3263.9 [2510.9 to 4242.8]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 1552.1 [1096.0 to 2198.2] | 2453.0 [1770.3 to 3399.0] | 2403.2 [1736.1 to 3326.7] | 2549.8 [1928.9 to 3370.5] | 2770.2 [2068.1 to 3710.6] | 3236.6 [2097.5 to 4994.4] | 2107.2 [1356.9 to 3272.5] | 1995.1 [1252.2 to 3178.7] | 1902.3 [1124.3 to 3219.0] | 2000.0 [1217.3 to 3286.1] | 2744.7 [1607.9 to 4685.1] | 2654.2 [1726.3 to 4080.8] | 2027.9 [1117.3 to 3680.5] | 2463.5 [1518.6 to 3996.3] | 2818.0 [2150.0 to 3693.6] | 2401.5 [1828.0 to 3155.0]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 1235.0 [853.9 to 1786.4] | 2217.1 [1542.4 to 3187.0] | 1987.9 [1402.9 to 2816.9] | 2012.2 [1493.1 to 2711.7] | 2032.1 [1439.1 to 2869.4] | 2218.4 [1463.1 to 3363.7] | 1998.1 [1258.7 to 3171.8] | 1943.4 [1217.9 to 3101.1] | 1824.1 [1074.4 to 3097.1] | 2355.2 [1414.7 to 3920.9] | 3247.7 [1958.8 to 5384.9] | 2270.8 [1442.0 to 3576.0] | 1985.3 [1110.9 to 3547.9] | 2335.7 [1355.9 to 4023.6] | 2538.8 [1942.3 to 3318.5] | 2007.4 [1569.1 to 2568.0]

31. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.1 in Two Dose Group.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.1.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
titer
  Day 1 | 249.7 [166.7 to 374.1]
  Day 15 | 4289.3 [2993.6 to 6145.7]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 3235.4 [2275.0 to 4601.3]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 2322.2 [1628.0 to 3312.5]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 4111.6 [3062.5 to 5520.2]
  Day 147 | 2616.7 [1867.5 to 3666.4]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 2088.0 [1490.7 to 2924.7]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 2006.1 [1382.0 to 2911.9]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 2136.6 [1418.6 to 3218.0]

32. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.2.12.1 in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.2.12.1.
Time Frame: Day 1 Pre-Booster Dose, Day 15
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
titer
  Day 1 | 173.5 [92.9 to 323.7] | 209.1 [105.8 to 413.0] | 217.0 [107.5 to 438.2] | 352.9 [193.9 to 642.6] | 345.2 [186.7 to 638.3]
  Day 15 | 1879.9 [1232.3 to 2868.0] | 1952.8 [1081.1 to 3527.3] | 2569.9 [1529.1 to 4319.2] | 3181.1 [2028.8 to 4987.9] | 2986.1 [1921.3 to 4641.2]

33. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.4/BA.5 in One Dose Groups.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.4/BA.5.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
titer
  Day 1 | 155.3 [108.9 to 221.5] | 170.8 [121.3 to 240.7] | 152.0 [108.0 to 213.9] | 195.4 [136.7 to 279.3] | 174.0 [119.5 to 253.3] | 206.8 [124.0 to 344.8] | 155.3 [94.3 to 255.9] | 183.7 [113.2 to 298.1] | 148.6 [91.5 to 241.3] | 150.1 [90.2 to 249.6] | 184.0 [106.9 to 316.9] | 257.6 [141.6 to 468.6] | 195.6 [108.1 to 353.9] | 254.8 [143.0 to 454.1] | 768.6 [565.0 to 1045.6] | 735.1 [533.9 to 1012.2]
  Day 15: number analyzed (Participants) | 27 | 25 | 26 | 25 | 26 | 0 | 0 | 0 | 1 | 0 | 0 | 46 | 49 | 50 | 100 | 100
  Day 15 | 1214.7 [815.9 to 1808.5] | 1349.8 [760.2 to 2396.8] | 1812.1 [1063.8 to 3086.9] | 2036.2 [1302.5 to 3183.2] | 1832.5 [1082.9 to 3100.8] |  |  |  | 169.0 [NA to NA] — 95% confidence interval was not estimable as data from only 1 participant was analyzed |  |  | 767.3 [474.6 to 1240.3] | 1084.3 [711.8 to 1651.9] | 1144.8 [766.8 to 1709.4] | 3577.0 [2894.3 to 4420.7] | 5906.9 [4617.4 to 7556.6]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 1035.7 [755.2 to 1420.4] | 1766.3 [1322.1 to 2359.8] | 1850.9 [1331.7 to 2572.7] | 1631.5 [1237.3 to 2151.3] | 1665.5 [1234.7 to 2246.6] | 870.9 [590.4 to 1284.6] | 1303.8 [899.6 to 1889.6] | 1754.5 [1181.4 to 2605.5] | 1397.6 [943.6 to 2070.0] | 1458.4 [1009.7 to 2106.6] | 1680.7 [1063.5 to 2656.0] | 948.1 [599.9 to 1498.5] | 1274.8 [799.1 to 2033.7] | 1463.9 [977.7 to 2191.8] | 3104.8 [2511.5 to 3838.3] | 4881.1 [3817.9 to 6240.5]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 756.3 [523.6 to 1092.5] | 1503.2 [1093.9 to 2065.6] | 1367.4 [962.2 to 1943.3] | 1297.3 [931.0 to 1807.7] | 1363.4 [987.9 to 1881.5] | 785.8 [475.4 to 1298.9] | 1032.5 [667.5 to 1597.2] | 1221.7 [744.6 to 2004.5] | 950.7 [535.5 to 1687.9] | 1021.8 [643.4 to 1622.7] | 1313.7 [795.7 to 2168.8] | 830.6 [493.5 to 1398.1] | 1201.3 [776.7 to 1858.2] | 1247.7 [763.0 to 2040.5] | 2163.2 [1676.3 to 2791.4] | 3774.7 [2960.5 to 4812.8]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 538.3 [354.5 to 817.4] | 1028.3 [714.5 to 1479.7] | 801.2 [547.5 to 1172.6] | 1037.4 [742.2 to 1450.1] | 1117.8 [788.8 to 1584.1] | 1327.5 [732.8 to 2405.1] | 707.8 [429.4 to 1166.5] | 971.0 [591.3 to 1594.5] | 868.4 [510.5 to 1477.3] | 824.6 [470.9 to 1444.1] | 1199.9 [694.2 to 2074.0] | 1460.0 [863.8 to 2467.5] | 1805.7 [1074.1 to 3035.6] | 1765.8 [1099.0 to 2837.2] | 2099.7 [1620.5 to 2720.5] | 3189.2 [2416.9 to 4208.3]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 1437.9 [981.0 to 2107.5] | 1951.1 [1399.6 to 2719.9] | 1733.1 [1237.6 to 2426.9] | 1950.2 [1412.5 to 2692.5] | 2023.5 [1469.2 to 2786.8] | 2655.1 [1512.9 to 4659.5] | 1451.4 [906.8 to 2323.1] | 1290.0 [808.6 to 2058.2] | 1620.4 [896.6 to 2928.6] | 1468.9 [838.9 to 2572.0] | 1727.2 [980.4 to 3042.8] | 2211.5 [1401.5 to 3489.8] | 1670.7 [976.1 to 2859.7] | 2263.3 [1433.7 to 3572.9] | 1843.8 [1416.4 to 2400.0] | 2419.0 [1826.0 to 3204.5]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 1208.4 [820.2 to 1780.3] | 1793.9 [1225.3 to 2626.4] | 1567.6 [1108.1 to 2217.8] | 1633.8 [1173.1 to 2275.3] | 1472.2 [1007.8 to 2150.5] | 2378.5 [1393.3 to 4060.6] | 1378.2 [846.0 to 2245.2] | 1180.6 [721.1 to 1932.9] | 1628.2 [899.4 to 2947.7] | 1972.5 [1163.4 to 3344.0] | 2122.8 [1179.5 to 3820.7] | 1993.5 [1208.8 to 3287.5] | 1628.0 [915.4 to 2895.1] | 2319.4 [1376.1 to 3909.6] | 1770.2 [1375.9 to 2277.6] | 2041.4 [1568.2 to 2657.3]

34. Primary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.4/BA.5 in Two Dose Group.
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against BA.4/BA.5.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
titer
  Day 1 | 132.1 [90.2 to 193.5]
  Day 15: number analyzed (Participants) | 1
  Day 15 | 816.0 [NA to NA] — 95% confidence interval is not estimable as data from only 1 participant was analyzed.
  Day 29: number analyzed (Participants) | 85
  Day 29 | 1416.8 [1004.5 to 1998.3]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 1148.9 [828.8 to 1592.6]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 2029.1 [1533.2 to 2685.4]
  Day 147 | 1195.3 [832.1 to 1716.9]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 1407.5 [963.9 to 2055.2]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 1419.5 [949.1 to 2123.1]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 1569.2 [1016.0 to 2423.6]

35. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against B.1.351 in One Dose Groups.
Description: GMR to D614G variant of Pseudovirus Neutralization Against B.1.351. GMR is calculated by dividing by the neutralization against D614G. The geometric mean of the ratio is then reported.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
ratio
  Day 1 | 0.25 [0.21 to 0.29] | 0.27 [0.22 to 0.33] | 0.24 [0.21 to 0.29] | 0.24 [0.20 to 0.29] | 0.27 [0.23 to 0.31] | 0.26 [0.20 to 0.32] | 0.28 [0.22 to 0.36] | 0.23 [0.18 to 0.29] | 0.26 [0.21 to 0.33] | 0.27 [0.21 to 0.33] | 0.23 [0.17 to 0.30] | 0.27 [0.21 to 0.37] | 0.25 [0.19 to 0.34] | 0.29 [0.21 to 0.39] | 0.38 [0.34 to 0.42] | 0.37 [0.32 to 0.42]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 0.36 [0.33 to 0.41] | 0.62 [0.57 to 0.68] | 0.41 [0.36 to 0.46] | 0.58 [0.50 to 0.68] | 0.41 [0.35 to 0.49] | 0.35 [0.30 to 0.42] | 0.57 [0.50 to 0.64] | 0.56 [0.49 to 0.64] | 0.55 [0.48 to 0.64] | 0.44 [0.39 to 0.50] | 0.40 [0.33 to 0.48] | 0.35 [0.30 to 0.41] | 0.53 [0.47 to 0.59] | 0.51 [0.45 to 0.57] | 0.56 [0.52 to 0.61] | 0.57 [0.52 to 0.62]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 0.30 [0.25 to 0.36] | 0.58 [0.53 to 0.63] | 0.38 [0.33 to 0.43] | 0.53 [0.44 to 0.63] | 0.38 [0.32 to 0.46] | 0.32 [0.27 to 0.38] | 0.50 [0.38 to 0.66] | 0.56 [0.49 to 0.64] | 0.57 [0.50 to 0.66] | 0.41 [0.36 to 0.46] | 0.38 [0.32 to 0.46] | 0.39 [0.33 to 0.47] | 0.60 [0.52 to 0.69] | 0.55 [0.48 to 0.62] | 0.43 [0.39 to 0.48] | 0.45 [0.40 to 0.49]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 0.31 [0.27 to 0.35] | 0.49 [0.44 to 0.54] | 0.34 [0.30 to 0.39] | 0.47 [0.40 to 0.55] | 0.39 [0.34 to 0.45] | 0.31 [0.25 to 0.38] | 0.53 [0.46 to 0.60] | 0.51 [0.44 to 0.58] | 0.54 [0.47 to 0.62] | 0.43 [0.38 to 0.48] | 0.43 [0.35 to 0.51] | 0.37 [0.31 to 0.43] | 0.54 [0.47 to 0.63] | 0.49 [0.43 to 0.56] | 0.42 [0.38 to 0.46] | 0.41 [0.36 to 0.46]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 0.29 [0.26 to 0.34] | 0.46 [0.39 to 0.54] | 0.31 [0.26 to 0.39] | 0.44 [0.40 to 0.49] | 0.40 [0.33 to 0.49] | 0.32 [0.27 to 0.38] | 0.41 [0.36 to 0.48] | 0.36 [0.30 to 0.43] | 0.40 [0.34 to 0.46] | 0.31 [0.25 to 0.37] | 0.32 [0.25 to 0.42] | 0.33 [0.29 to 0.39] | 0.47 [0.41 to 0.54] | 0.46 [0.40 to 0.52] | 0.50 [0.44 to 0.57] | 0.49 [0.43 to 0.55]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 0.30 [0.25 to 0.36] | 0.39 [0.33 to 0.47] | 0.31 [0.26 to 0.38] | 0.37 [0.31 to 0.44] | 0.37 [0.33 to 0.42] | 0.45 [0.38 to 0.55] | 0.53 [0.46 to 0.62] | 0.43 [0.35 to 0.54] | 0.47 [0.40 to 0.54] | 0.47 [0.41 to 0.55] | 0.49 [0.41 to 0.59] | 0.47 [0.40 to 0.55] | 0.60 [0.51 to 0.71] | 0.55 [0.46 to 0.65] | 0.37 [0.33 to 0.41] | 0.34 [0.31 to 0.38]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 0.33 [0.28 to 0.38] | 0.43 [0.39 to 0.48] | 0.33 [0.27 to 0.40] | 0.39 [0.34 to 0.45] | 0.36 [0.30 to 0.43] | 0.36 [0.30 to 0.43] | 0.42 [0.35 to 0.50] | 0.36 [0.30 to 0.42] | 0.42 [0.36 to 0.49] | 0.32 [0.27 to 0.38] | 0.35 [0.29 to 0.42] | 0.34 [0.28 to 0.40] | 0.36 [0.25 to 0.52] | 0.37 [0.32 to 0.44] | 0.48 [0.43 to 0.54] | 0.47 [0.42 to 0.53]

36. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against B.1.351 in Two Dose Group.
Description: as for outcome 35
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
ratio
  Day 1 | 0.25 [0.21 to 0.31]
  Day 15 | 0.63 [0.57 to 0.69]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 0.61 [0.55 to 0.67]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 0.54 [0.49 to 0.60]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 0.63 [0.58 to 0.69]
  Day 147 | 0.51 [0.46 to 0.56]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 0.44 [0.37 to 0.53]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 0.48 [0.41 to 0.58]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 0.37 [0.31 to 0.44]

37. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against B.1.617.2 in One Dose Groups.
Description: GMR to D614G variant of Pseudovirus Neutralization Against B.1.617.2. GMR is calculated by dividing by the neutralization against D614G. The geometric mean of the ratio is then reported.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
ratio
  Day 1 | 0.49 [0.45 to 0.54] | 0.47 [0.42 to 0.51] | 0.50 [0.47 to 0.54] | 0.49 [0.46 to 0.53] | 0.49 [0.46 to 0.53] | 0.47 [0.42 to 0.54] | 0.47 [0.40 to 0.55] | 0.45 [0.39 to 0.51] | 0.50 [0.45 to 0.55] | 0.50 [0.45 to 0.56] | 0.43 [0.38 to 0.49] | 0.52 [0.47 to 0.57] | 0.51 [0.46 to 0.57] | 0.46 [0.35 to 0.60] | 0.45 [0.42 to 0.48] | 0.47 [0.44 to 0.50]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 0.55 [0.52 to 0.58] | 0.62 [0.59 to 0.66] | 0.60 [0.56 to 0.64] | 0.60 [0.57 to 0.64] | 0.53 [0.46 to 0.62] | 0.50 [0.46 to 0.55] | 0.58 [0.53 to 0.63] | 0.55 [0.49 to 0.62] | 0.50 [0.46 to 0.55] | 0.53 [0.50 to 0.58] | 0.47 [0.41 to 0.54] | 0.45 [0.42 to 0.49] | 0.52 [0.49 to 0.55] | 0.48 [0.45 to 0.52] | 0.53 [0.51 to 0.55] | 0.54 [0.52 to 0.56]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 0.49 [0.46 to 0.53] | 0.58 [0.54 to 0.62] | 0.60 [0.57 to 0.64] | 0.57 [0.54 to 0.61] | 0.55 [0.51 to 0.59] | 0.51 [0.47 to 0.56] | 0.57 [0.53 to 0.63] | 0.55 [0.49 to 0.62] | 0.58 [0.52 to 0.64] | 0.55 [0.50 to 0.59] | 0.49 [0.45 to 0.53] | 0.56 [0.52 to 0.59] | 0.63 [0.58 to 0.68] | 0.60 [0.56 to 0.64] | 0.43 [0.40 to 0.45] | 0.45 [0.42 to 0.48]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 0.46 [0.43 to 0.49] | 0.55 [0.52 to 0.59] | 0.50 [0.47 to 0.53] | 0.51 [0.44 to 0.58] | 0.52 [0.49 to 0.56] | 0.55 [0.50 to 0.60] | 0.59 [0.55 to 0.64] | 0.60 [0.54 to 0.66] | 0.56 [0.52 to 0.61] | 0.54 [0.50 to 0.59] | 0.54 [0.49 to 0.60] | 0.48 [0.45 to 0.52] | 0.57 [0.52 to 0.61] | 0.54 [0.50 to 0.59] | 0.43 [0.41 to 0.46] | 0.43 [0.41 to 0.46]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 0.42 [0.40 to 0.45] | 0.47 [0.41 to 0.54] | 0.43 [0.37 to 0.50] | 0.46 [0.43 to 0.49] | 0.42 [0.36 to 0.48] | 0.44 [0.40 to 0.48] | 0.44 [0.40 to 0.48] | 0.46 [0.42 to 0.50] | 0.42 [0.38 to 0.46] | 0.44 [0.41 to 0.48] | 0.37 [0.31 to 0.45] | 0.39 [0.36 to 0.43] | 0.52 [0.47 to 0.57] | 0.47 [0.43 to 0.51] | 0.51 [0.48 to 0.54] | 0.55 [0.52 to 0.59]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 0.42 [0.39 to 0.46] | 0.41 [0.36 to 0.48] | 0.40 [0.34 to 0.46] | 0.42 [0.39 to 0.45] | 0.42 [0.39 to 0.45] | 0.48 [0.44 to 0.54] | 0.47 [0.43 to 0.52] | 0.47 [0.40 to 0.54] | 0.45 [0.40 to 0.50] | 0.50 [0.46 to 0.55] | 0.48 [0.43 to 0.53] | 0.50 [0.45 to 0.55] | 0.56 [0.50 to 0.62] | 0.50 [0.46 to 0.55] | 0.47 [0.44 to 0.50] | 0.47 [0.44 to 0.51]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 0.46 [0.42 to 0.49] | 0.49 [0.45 to 0.54] | 0.47 [0.40 to 0.55] | 0.46 [0.42 to 0.50] | 0.43 [0.37 to 0.50] | 0.48 [0.43 to 0.54] | 0.48 [0.43 to 0.54] | 0.47 [0.41 to 0.55] | 0.47 [0.41 to 0.53] | 0.46 [0.41 to 0.53] | 0.46 [0.41 to 0.52] | 0.40 [0.36 to 0.45] | 0.41 [0.29 to 0.58] | 0.45 [0.41 to 0.49] | 0.64 [0.60 to 0.68] | 0.68 [0.63 to 0.72]

38. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against B.1.617.2 in Two Dose Group.
Description: as for outcome 37
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
ratio
  Day 1 | 0.45 [0.38 to 0.53]
  Day 15 | 0.56 [0.47 to 0.67]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 0.58 [0.55 to 0.62]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 0.56 [0.53 to 0.60]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 0.60 [0.57 to 0.64]
  Day 147 | 0.50 [0.43 to 0.58]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 0.41 [0.35 to 0.48]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 0.44 [0.37 to 0.51]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 0.39 [0.33 to 0.45]

39. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against BA.1 in One Dose Groups.
Description: GMR to D614G variant of Pseudovirus Neutralization Against BA.1. GMR is calculated by dividing by the neutralization against D614G. The geometric mean of the ratio is then reported.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
ratio
  Day 1 | 0.08 [0.07 to 0.10] | 0.08 [0.07 to 0.09] | 0.08 [0.06 to 0.10] | 0.09 [0.07 to 0.11] | 0.10 [0.08 to 0.12] | 0.09 [0.07 to 0.12] | 0.08 [0.06 to 0.11] | 0.08 [0.06 to 0.11] | 0.07 [0.05 to 0.10] | 0.08 [0.06 to 0.11] | 0.07 [0.05 to 0.11] | 0.08 [0.06 to 0.11] | 0.08 [0.06 to 0.12] | 0.07 [0.05 to 0.09] | 0.15 [0.13 to 0.17] | 0.13 [0.11 to 0.16]
  Day 15: number analyzed (Participants) | 99 | 112 | 101 | 99 | 97 | 47 | 51 | 53 | 51 | 51 | 52 | 46 | 49 | 50 | 100 | 100
  Day 15 | 0.13 [0.11 to 0.15] | 0.25 [0.21 to 0.29] | 0.19 [0.16 to 0.22] | 0.31 [0.27 to 0.36] | 0.20 [0.17 to 0.24] | 0.12 [0.10 to 0.16] | 0.25 [0.21 to 0.30] | 0.30 [0.26 to 0.35] | 0.18 [0.15 to 0.21] | 0.16 [0.13 to 0.19] | 0.20 [0.16 to 0.24] | 0.15 [0.12 to 0.19] | 0.20 [0.15 to 0.27] | 0.16 [0.12 to 0.22] | 0.24 [0.21 to 0.27] | 0.19 [0.16 to 0.23]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 97 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 0.12 [0.10 to 0.14] | 0.24 [0.20 to 0.28] | 0.18 [0.15 to 0.22] | 0.28 [0.24 to 0.33] | 0.20 [0.16 to 0.24] | 0.10 [0.08 to 0.12] | 0.16 [0.12 to 0.21] | 0.25 [0.21 to 0.29] | 0.15 [0.12 to 0.18] | 0.13 [0.11 to 0.16] | 0.14 [0.11 to 0.17] | 0.10 [0.07 to 0.14] | 0.17 [0.11 to 0.26] | 0.12 [0.09 to 0.17] | 0.17 [0.14 to 0.19] | 0.14 [0.11 to 0.17]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 0.09 [0.08 to 0.11] | 0.17 [0.15 to 0.20] | 0.13 [0.11 to 0.16] | 0.17 [0.14 to 0.20] | 0.15 [0.12 to 0.19] | 0.14 [0.11 to 0.18] | 0.26 [0.21 to 0.32] | 0.37 [0.31 to 0.43] | 0.21 [0.17 to 0.25] | 0.19 [0.15 to 0.23] | 0.24 [0.18 to 0.31] | 0.11 [0.09 to 0.14] | 0.14 [0.09 to 0.22] | 0.12 [0.09 to 0.17] | 0.27 [0.24 to 0.30] | 0.21 [0.18 to 0.24]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 0.11 [0.09 to 0.13] | 0.21 [0.18 to 0.25] | 0.14 [0.11 to 0.17] | 0.21 [0.18 to 0.25] | 0.17 [0.14 to 0.21] | 0.14 [0.11 to 0.18] | 0.19 [0.14 to 0.26] | 0.25 [0.21 to 0.31] | 0.16 [0.13 to 0.21] | 0.16 [0.12 to 0.20] | 0.18 [0.13 to 0.25] | 0.15 [0.12 to 0.19] | 0.25 [0.19 to 0.32] | 0.17 [0.14 to 0.22] | 0.29 [0.26 to 0.33] | 0.26 [0.23 to 0.30]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 0.14 [0.11 to 0.16] | 0.19 [0.16 to 0.23] | 0.19 [0.16 to 0.23] | 0.21 [0.18 to 0.25] | 0.22 [0.19 to 0.25] | 0.21 [0.16 to 0.27] | 0.27 [0.23 to 0.32] | 0.28 [0.21 to 0.37] | 0.18 [0.14 to 0.23] | 0.21 [0.17 to 0.26] | 0.26 [0.20 to 0.32] | 0.21 [0.17 to 0.26] | 0.19 [0.11 to 0.32] | 0.19 [0.14 to 0.25] | 0.29 [0.25 to 0.33] | 0.23 [0.20 to 0.26]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 0.14 [0.11 to 0.18] | 0.25 [0.22 to 0.30] | 0.23 [0.19 to 0.28] | 0.25 [0.21 to 0.29] | 0.21 [0.17 to 0.25] | 0.17 [0.13 to 0.21] | 0.26 [0.21 to 0.32] | 0.29 [0.24 to 0.36] | 0.19 [0.15 to 0.24] | 0.19 [0.15 to 0.25] | 0.26 [0.21 to 0.32] | 0.17 [0.13 to 0.22] | 0.19 [0.11 to 0.32] | 0.16 [0.12 to 0.22] | 0.30 [0.27 to 0.34] | 0.24 [0.20 to 0.27]

40. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against BA.1 in Two Dose Group.
Description: as for outcome 39
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
ratio
  Day 1 | 0.07 [0.06 to 0.10]
  Day 15 | 0.24 [0.20 to 0.29]
  Day 29: number analyzed (Participants) | 85
  Day 29 | 0.25 [0.22 to 0.29]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 0.21 [0.17 to 0.25]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 0.25 [0.22 to 0.29]
  Day 147 | 0.26 [0.22 to 0.32]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 0.17 [0.14 to 0.21]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 0.23 [0.19 to 0.28]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 0.21 [0.17 to 0.26]

41. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against BA.2.12.1 in One Dose Groups.
Description: GMR to D614G variant of Pseudovirus Neutralization Against BA.2.12.1. GMR is calculated by dividing by the neutralization against D614G. The geometric mean of the ratio is then reported.
Time Frame: Day 1 Pre-Booster Dose, Day 15
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ratio
  Day 1 | 0.07 [0.05 to 0.10] | 0.04 [0.03 to 0.06] | 0.05 [0.03 to 0.09] | 0.06 [0.04 to 0.08] | 0.07 [0.05 to 0.10]
  Day 15 | 0.11 [0.08 to 0.15] | 0.13 [0.09 to 0.20] | 0.12 [0.09 to 0.16] | 0.18 [0.14 to 0.22] | 0.14 [0.11 to 0.18]

42. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against BA.4/BA.5 in One Dose Groups.
Description: GMR to D614G variant of Pseudovirus Neutralization Against BA.4/BA.5. GMR is calculated by dividing by the neutralization against D614G. The geometric mean of the ratio is then reported.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 271, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 101 | 99 | 97 | 49 | 52 | 54 | 51 | 52 | 53 | 48 | 49 | 52 | 100 | 100
ratio
  Day 1 | 0.05 [0.04 to 0.06] | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.06] | 0.05 [0.04 to 0.06] | 0.04 [0.04 to 0.06] | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.06] | 0.04 [0.03 to 0.06] | 0.03 [0.03 to 0.05] | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.07] | 0.06 [0.04 to 0.08] | 0.05 [0.03 to 0.06] | 0.10 [0.09 to 0.12] | 0.09 [0.08 to 0.11]
  Day 15: number analyzed (Participants) | 27 | 25 | 26 | 25 | 26 | 0 | 0 | 0 | 1 | 0 | 0 | 46 | 49 | 50 | 100 | 100
  Day 15 | 0.07 [0.06 to 0.09] | 0.09 [0.06 to 0.13] | 0.08 [0.06 to 0.11] | 0.11 [0.10 to 0.14] | 0.09 [0.06 to 0.12] |  |  |  | 0.11 [NA to NA] — 95% confidence interval is not estimable as data from only 1 participant was analyzed. |  |  | 0.09 [0.07 to 0.12] | 0.11 [0.08 to 0.16] | 0.11 [0.09 to 0.15] | 0.13 [0.11 to 0.15] | 0.18 [0.15 to 0.21]
  Day 29: number analyzed (Participants) | 97 | 113 | 100 | 98 | 95 | 49 | 52 | 52 | 51 | 52 | 52 | 48 | 46 | 51 | 99 | 98
  Day 29 | 0.06 [0.05 to 0.08] | 0.11 [0.09 to 0.13] | 0.10 [0.08 to 0.13] | 0.11 [0.09 to 0.14] | 0.09 [0.08 to 0.11] | 0.05 [0.04 to 0.07] | 0.08 [0.06 to 0.11] | 0.11 [0.09 to 0.14] | 0.09 [0.07 to 0.11] | 0.07 [0.06 to 0.09] | 0.07 [0.05 to 0.09] | 0.09 [0.07 to 0.12] | 0.09 [0.06 to 0.14] | 0.10 [0.08 to 0.13] | 0.10 [0.09 to 0.11] | 0.13 [0.11 to 0.16]
  Day 91: number analyzed (Participants) | 94 | 111 | 99 | 98 | 96 | 48 | 50 | 51 | 50 | 51 | 51 | 48 | 48 | 51 | 98 | 98
  Day 91 | 0.06 [0.05 to 0.08] | 0.10 [0.09 to 0.13] | 0.08 [0.07 to 0.10] | 0.09 [0.07 to 0.11] | 0.08 [0.07 to 0.10] | 0.09 [0.06 to 0.12] | 0.14 [0.12 to 0.18] | 0.15 [0.11 to 0.20] | 0.11 [0.09 to 0.15] | 0.10 [0.08 to 0.13] | 0.11 [0.08 to 0.16] | 0.07 [0.05 to 0.10] | 0.10 [0.06 to 0.14] | 0.10 [0.08 to 0.14] | 0.15 [0.13 to 0.17] | 0.20 [0.17 to 0.23]
  Day 181: number analyzed (Participants) | 93 | 107 | 97 | 96 | 94 | 42 | 49 | 47 | 50 | 50 | 47 | 46 | 43 | 50 | 94 | 95
  Day 181 | 0.08 [0.06 to 0.10] | 0.14 [0.11 to 0.16] | 0.09 [0.07 to 0.11] | 0.14 [0.11 to 0.16] | 0.11 [0.09 to 0.14] | 0.10 [0.07 to 0.15] | 0.11 [0.08 to 0.15] | 0.13 [0.10 to 0.17] | 0.11 [0.08 to 0.14] | 0.09 [0.06 to 0.13] | 0.11 [0.08 to 0.15] | 0.12 [0.09 to 0.15] | 0.18 [0.14 to 0.23] | 0.13 [0.10 to 0.17] | 0.18 [0.16 to 0.21] | 0.26 [0.22 to 0.30]
  Day 271: number analyzed (Participants) | 90 | 101 | 92 | 96 | 89 | 41 | 49 | 49 | 47 | 48 | 50 | 46 | 43 | 47 | 89 | 94
  Day 271 | 0.13 [0.10 to 0.15] | 0.15 [0.13 to 0.18] | 0.14 [0.11 to 0.17] | 0.16 [0.14 to 0.20] | 0.16 [0.14 to 0.19] | 0.17 [0.12 to 0.23] | 0.19 [0.15 to 0.23] | 0.18 [0.14 to 0.23] | 0.15 [0.12 to 0.20] | 0.15 [0.12 to 0.20] | 0.16 [0.12 to 0.21] | 0.18 [0.14 to 0.21] | 0.16 [0.10 to 0.25] | 0.17 [0.14 to 0.21] | 0.19 [0.17 to 0.21] | 0.23 [0.20 to 0.27]
  Day 366: number analyzed (Participants) | 90 | 101 | 95 | 95 | 91 | 44 | 48 | 49 | 48 | 47 | 48 | 46 | 40 | 45 | 89 | 90
  Day 366 | 0.14 [0.11 to 0.18] | 0.20 [0.17 to 0.25] | 0.18 [0.15 to 0.22] | 0.20 [0.17 to 0.24] | 0.15 [0.12 to 0.19] | 0.18 [0.13 to 0.24] | 0.18 [0.14 to 0.23] | 0.18 [0.13 to 0.23] | 0.17 [0.12 to 0.23] | 0.16 [0.13 to 0.21] | 0.17 [0.12 to 0.24] | 0.15 [0.12 to 0.19] | 0.16 [0.09 to 0.26] | 0.16 [0.13 to 0.20] | 0.21 [0.19 to 0.24] | 0.24 [0.21 to 0.28]

43. Primary Outcome: Geometric Mean Ratio (GMR) to D614G Variant of Pseudovirus Neutralization Against BA.4/BA.5 in Two Dose Group.
Description: as for outcome 42
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 57, Day 85, Day 147, Day 237, Day 327, Day 422
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses)
Number analyzed (Participants) | 86
ratio
  Day 1 | 0.04 [0.03 to 0.05]
  Day 15: number analyzed (Participants) | 1
  Day 15 | 0.06 [NA to NA] — 95% confidence interval was not estimable as data from only 1 participant was analyzed
  Day 29: number analyzed (Participants) | 85
  Day 29 | 0.11 [0.09 to 0.13]
  Day 57: number analyzed (Participants) | 84
  Day 57 | 0.10 [0.09 to 0.12]
  Day 85: number analyzed (Participants) | 85
  Day 85 | 0.12 [0.11 to 0.14]
  Day 147 | 0.12 [0.10 to 0.15]
  Day 237: number analyzed (Participants) | 85
  Day 237 | 0.12 [0.09 to 0.14]
  Day 327: number analyzed (Participants) | 84
  Day 327 | 0.16 [0.13 to 0.20]
  Day 422: number analyzed (Participants) | 82
  Day 422 | 0.15 [0.12 to 0.20]

44. Secondary Outcome: Frequency of Any Adverse Events (AEs) Leading to Withdrawal From the Study.
Description: Number of participants that experienced any AE during the course of the study that resulted in withdrawal from the study.
Time Frame: Day 1 to study completion (through up to Day 366) for Arms 1,2,4,5,6,7,8,9,10,11,12,13,14,15,16,17 and Day 1 to study completion (through up to Day 422) for Arm 3.
Population: The Safety Analysis population for the study includes all participants who received at least one dose of vaccine. Participants in Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) who did not receive second dose were analyzed as part of Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

45. Secondary Outcome: Frequency of Any Adverse Events of Special Interest (AESIs)
Description: Number of participants that experienced any AESI during the course of the study.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 3 | 7 | 7 | 5 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 2

46. Secondary Outcome: Frequency of Any Medically Attended Adverse Events (MAAEs)
Description: Number of participants that experienced any MAAE during the course of the study. Medically Attended Adverse Events (MAAEs) are defined as a hospitalization < 24 hours, emergency room visit or an otherwise unscheduled visit to or from medical personnel for any reason; and considered related or possibly related to study product
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Frequency of Any New Onset Chronic Medical Conditions (NOCMCs)
Description: Number of participants that experienced any NOCMC during the course of the study.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 2 | 8 | 4 | 5 | 3 | 1 | 2 | 5 | 5 | 0 | 1 | 0 | 1 | 2 | 1 | 5 | 2

48. Secondary Outcome: Frequency of Any Serious Adverse Events (SAEs)
Description: Number of participants that experienced any SAEs during the course of the study. An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 4 | 4 | 7 | 2 | 3 | 4 | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 1 | 1 | 0 | 0

49. Secondary Outcome: Frequency of Systemic Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any systemic solicited AEs through 7 days post any vaccination. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever.
Time Frame: Day 1 through Day 8 for Arms 1, 2, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14,15, 16, and 17 and through 7 days post any vaccination for Arm 3.
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 82 | 88 | 70 | 80 | 81 | 80 | 40 | 42 | 37 | 33 | 36 | 39 | 33 | 33 | 35 | 80 | 83

50. Secondary Outcome: Frequency of Local Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any local solicited AEs through 7 days post any vaccination. Local events include: Injection Site Pain, Injection site Erythema, and Injection site Edema/Induration.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 93 | 101 | 77 | 87 | 82 | 80 | 38 | 41 | 43 | 40 | 43 | 46 | 40 | 42 | 42 | 82 | 86

51. Secondary Outcome: Frequency of Any Unsolicited Adverse Events (AEs)
Description: Number of participants that experienced any Unsolicited AEs through 28 days post vaccination.
Time Frame: Day 1 through Day 29 for Arms 1, 2, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14,15, 16, and 17 and 28 days post any vaccination for Arm 3.
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
Number analyzed (Participants) | 99 | 113 | 86 | 101 | 99 | 99 | 50 | 52 | 54 | 51 | 52 | 53 | 49 | 51 | 52 | 101 | 101
Participants | 26 | 40 | 39 | 31 | 35 | 33 | 17 | 12 | 14 | 13 | 19 | 16 | 15 | 13 | 11 | 33 | 28

ADVERSE EVENTS:
Time Frame: Solicited AEs (i.e., reactogenicity) will be collected using a memory aid from the time of each vaccination through 7 days post each vaccination. Unsolicited AEs of all severities will be reported from the time of study product administration through 28 days post each vaccination. After 28 days post vaccination through Day 366 (Arms 1,2,4,5,6,7,8,9,10,11,12,13,14,15,16,17) or Day 422 (Arm 3) only AESIs/MAAEs/SAEs/NOCMCs and AEs leading to withdrawal were reported as AEs.
Description: Participants in Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) were included in Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) for reporting AEs that occurred after Dose 1 but before Dose 2.
Arm/Group | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype])
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/199 | 0/86 | 0/101 | 0/99 | 1/99 | 0/50 | 0/52 | 0/54 | 0/51 | 0/52 | 0/53 | 0/49 | 0/51 | 1/52 | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 4/99 | 4/199 | 6/86 | 2/101 | 3/99 | 2/99 | 0/50 | 0/52 | 1/54 | 1/51 | 5/52 | 1/53 | 1/49 | 1/51 | 1/52 | 0/101 | 0/101
Other Adverse Events (participants affected / at risk) | 98/99 | 185/199 | 76/86 | 98/101 | 94/99 | 89/99 | 46/50 | 47/52 | 49/54 | 42/51 | 48/52 | 51/53 | 42/49 | 46/51 | 49/52 | 96/101 | 94/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) (N=99) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) (N=199) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) (N=86) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) (N=101) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) (N=99) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) (N=99) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) (N=50) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) (N=52) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) (N=54) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) (N=51) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) (N=52) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) (N=53) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) (N=49) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) (N=51) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) (N=52) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) (N=101) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype]) (N=101)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Right upper lobe pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Worsening orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Traumatic lisfranc injury to right foot (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Right parietal hemorrhage stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Perforated duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Vasa previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Great toe cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Sickle cell crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Non reducible hemorrhoid (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Diastasis recti (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Reoccurring appendiceal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Enlargement of ovarian cysts (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Clot retention in the urinary bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Bleeding stomach ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Acute COVID19 multifocal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Ascending colon adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 - Arm 01 (Moderna mRNA1273 Prototype) (N=99) | Stage 1 - Arm 02 (Moderna mRNA 1273 Beta + Omicron - 1 Dose) (N=199) | Stage 1 - Arm 03 (Moderna mRNA 1273 Beta + Omicron - 2 Doses) (N=86) | Stage 1 - Arm 04 (Moderna mRNA1273 Delta + Omicron) (N=101) | Stage 1 - Arm 05 (Moderna mRNA1273 Omicron) (N=99) | Stage 1 - Arm 06 (Moderna mRNA1273 Omicron + Prototype) (N=99) | Stage 2 - Arm 07 (Pfizer/BNT BNT162b2 Wildtype [Prototype]) (N=50) | Stage 2 - Arm 08 (Pfizer/BNT BNT162b2 Beta + Omicron) (N=52) | Stage 2 - Arm 09 (Pfizer/BNT BNT162b2 Omicron) (N=54) | Stage 2 - Arm 10 (Pfizer/BNT BNT162b2 Beta) (N=51) | Stage 2 - Arm 11 (Pfizer/BNT BNT162b2 Beta + Wildtype [Prototype]) (N=52) | Stage 2 - Arm 12 (Pfizer/BNT BNT162b2 Omicron + Wildtype [Prototype]) (N=53) | Stage 3 - Arm 13 (Sanofi CoV2 preS dTM-AS03 Prototype) (N=49) | Stage 3 - Arm 14 (Sanofi CoV2 preS dTM-AS03 Beta) (N=51) | Stage 3 - Arm 15 (Sanofi CoV2 preS dTM-AS03 Beta + Prototype) (N=52) | Stage 4 - Arm 16 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.1 + Wildtype [Prototype]) (N=101) | Stage 4 - Arm 17 (Pfizer/BNT BNT162b2 Bivalent Omicron BA.4/BA.5 + Wildtype [Prototype]) (N=101)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (9)
Nausea (Gastrointestinal disorders) | 11 (11) | 36 (36) | 10 (10) | 10 (10) | 10 (10) | 28 (28) | 8 (8) | 6 (6) | 7 (7) | 7 (7) | 7 (7) | 1 (1) | 6 (6) | 5 (5) | 4 (4) | 15 (15) | 16 (16)
Chills (General disorders) | 32 (32) | 51 (51) | 17 (17) | 33 (33) | 29 (29) | 33 (33) | 8 (8) | 7 (7) | 11 (11) | 11 (11) | 9 (9) | 7 (7) | 9 (9) | 7 (7) | 9 (9) | 22 (22) | 34 (34)
Fatigue (General disorders) | 66 (66) | 128 (128) | 43 (43) | 68 (68) | 67 (67) | 71 (71) | 37 (37) | 32 (32) | 26 (26) | 29 (29) | 31 (31) | 31 (31) | 25 (25) | 23 (23) | 29 (29) | 65 (65) | 74 (74)
Pyrexia (General disorders) | 5 (5) | 14 (14) | 3 (3) | 13 (13) | 6 (6) | 12 (12) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 7 (7)
Vaccination site induration (General disorders) | 21 (21) | 53 (53) | 24 (24) | 20 (20) | 17 (17) | 20 (20) | 10 (10) | 5 (5) | 11 (11) | 12 (12) | 9 (9) | 11 (11) | 17 (17) | 11 (11) | 13 (13) | 19 (19) | 23 (23)
Vaccination site pain (General disorders) | 89 (89) | 168 (168) | 63 (63) | 83 (83) | 82 (82) | 76 (76) | 36 (36) | 40 (40) | 42 (42) | 38 (38) | 42 (42) | 44 (44) | 38 (38) | 37 (37) | 40 (40) | 81 (81) | 84 (84)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (24) | 49 (49) | 9 (9) | 26 (26) | 24 (24) | 24 (24) | 10 (10) | 16 (16) | 12 (12) | 10 (10) | 11 (11) | 7 (7) | 6 (6) | 6 (6) | 6 (6) | 20 (20) | 26 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 67 (67) | 105 (105) | 39 (39) | 49 (49) | 60 (60) | 64 (64) | 28 (28) | 30 (30) | 23 (23) | 23 (23) | 24 (24) | 25 (25) | 19 (19) | 20 (20) | 22 (22) | 51 (51) | 59 (59)
Headache (Nervous system disorders) | 33 (33) | 86 (86) | 27 (27) | 43 (43) | 39 (39) | 48 (48) | 26 (26) | 17 (17) | 20 (20) | 23 (23) | 19 (19) | 19 (19) | 22 (22) | 17 (17) | 14 (14) | 45 (45) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT05289037/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT05289037/SAP_002.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT05289037/ICF_000.pdf